CLINICAL TRIAL: NCT01571362
Title: A Multicenter, 12 Week, Double-blind, Placebo-controlled, Randomized Withdrawal Study To Determine The Efficacy And Safety Of Alo-02 (Oxycodone Hydrochloride And Naltrexone Hydrochloride) Extended-release Capsules In Subjects With Moderate To Severe Chronic Low Back Pain
Brief Title: A Research Study of an Investigational Drug ALO-02 (Oxycodone Hydrochloride and Naltrexone Hydrochloride) in Patients With Moderate to Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B4531002; B4531002; ALO-02-10-3002 (Other: Alias Study Number)
Record Dates: First submitted 2012-04-03; First posted 2012-04-05 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Chronic Pain; Low Back Pain; Analgesia
Keywords: oxycodone; naltrexone; chronic pain; low back pain
MeSH Terms: conditions — Chronic Pain; Low Back Pain; Agnosia | interventions — oxycodone naltrexone combination; Oxycodone; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALO-02 (Experimental)
  Interventions: Drug: ALO-02
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALO-02 — 20 to 160mg total daily dose of oxycodone, divided into symmetric doses and administered twice daily
  Other Names: oxycodone HCl and naltrexone HCl
  Arms: ALO-02
Drug: Placebo — oral placebo, divided into symmetric doses and administered twice daily
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the analgesic efficacy and safety of ALO-02 extended-release capsules, when compared to placebo, in subjects with moderate to severe chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe chronic low back pain present for at least 3 months.
* Require a continuous around-the-clock opioid analgesic for an extended period of time.
* Refrain from taking other opioid and non-opioid medications during the study.

Exclusion Criteria:

* Active or within a past 2 years a history of lumbosacral radiculopathy or chronic low back pain due to other underlying disorders such as spinal stenosis with neurologic impairment, cancer, infection, or post-surgical intervention.
* Documented diagnosis of ongoing pain due to other chronic pain conditions which may interfere with assessment of chronic low back pain.
* Active or ongoing or history of alcohol or drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (52):
  - Coastal Clinical Research, Inc., Mobile, Alabama
  - Dedicated Clinical Research, Goodyear, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Premier Research Group Limited, Phoenix, Arizona
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Med Center, Carmichael, California
  - Med Investigations, Inc., Fair Oaks, California
  - Neuro-Pain Medical Center, Fresno, California
  - Pacific Coast Pain Management Center, Laguna Hills, California
  - Long Beach Center for Clinical Research - previous addresse, Long Beach, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Providence Clinical Research, North Hollywood, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Lynn Institute of the Rockies Medical Centre, Colorado Springs, Colorado
  - Avail Clinical Research, LLC, DeLand, Florida
  - Ormond Medical Arts pharmaceutical Research Center, Ormond Beach, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - The Office of Martin E. Hale, MD, PA, Plantation, Florida
  - Accord Clinical Research, LLC- Duplicate 2, Port Orange, Florida
  - Accord Clinical Research, LLC- Duplicate, Port Orange, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Drug Studies America, Marietta, Georgia
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Mid-Atlantic Medical Research - Research Department, Hollywood, Maryland
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Mercy Health Research, St Louis, Missouri
  - Heartland Clinical Research, Inc., Omaha, Nebraska
  - Office of Stephen H. Miller, M.D., Las Vegas, Nevada
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Drug Trials America, Hartsdale, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Research Across America, New York, New York
  - Upstate Clinical Research Associates, LLC, Williamsville, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Community Research, Cincinnati, Ohio
  - Columbus Clinical Research, Columbus, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Associated Orthopedics, Oklahoma City, Oklahoma
  - Hillcrest Clinical Research, Oklahoma City, Oklahoma
  - Allegheny Pain Management, PC, Altoona, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Pain Research of Charleston, Charleston, South Carolina
  - TLM Medical Services, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - KRK Medical Research, Dallas, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Quality Research Inc., San Antonio, Texas
  - Lee Medical Associates, San Antonio, Texas
  - Progressive Clinical Research, P.A., San Antonio, Texas

REFERENCES:
- [Derived] Gimbel JS, Rauck RL, Bass A, Wilson J, Pixton G, Malhotra B, Wilson G, Wolfram G. Effects of naltrexone exposure observed in two phase three studies with ALO-02, an extended-release oxycodone surrounding sequestered naltrexone. J Opioid Manag. 2019 Sep/Oct;15(5):417-427. doi: 10.5055/jom.2019.0530. PMID 31849032
- [Derived] Wilson JG, Bass A, Pixton GC, Wolfram G, Rauck RL. Safety and tolerability of ALO-02 (oxycodone hydrochloride and sequestered naltrexone hydrochloride) extended-release capsules in older patients: a pooled analysis of two clinical trials. Curr Med Res Opin. 2020 Jan;36(1):91-99. doi: 10.1080/03007995.2019.1661679. Epub 2019 Sep 17. PMID 31456431
- [Derived] Weil AJ, Masters ET, Barsdorf AI, Bass A, Pixton G, Wilson JG, Wolfram G. Patient-reported health-related quality of life, work productivity, and activity impairment during treatment with ALO-02 (extended-release oxycodone and sequestered naltrexone) for moderate-to-severe chronic low back pain. Health Qual Life Outcomes. 2017 Oct 17;15(1):202. doi: 10.1186/s12955-017-0749-y. PMID 29041942
- [Derived] Rauck RL, Hale ME, Bass A, Bramson C, Pixton G, Wilson JG, Setnik B, Meisner P, Sommerville KW, Malhotra BK, Wolfram G. A randomized double-blind, placebo-controlled efficacy and safety study of ALO-02 (extended-release oxycodone surrounding sequestered naltrexone) for moderate-to-severe chronic low back pain treatment. Pain. 2015 Sep;156(9):1660-1669. doi: 10.1097/j.pain.0000000000000230. PMID 25993547
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4531002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Double-Blind, Placebo-Controlled, Randomized Withdrawal Study to Determine the Efficacy and Safety of ALO-02 Extended-Release Capsules in participants with Moderate to Severe Chronic Low Back Pain
Pre-assignment Details: A total of 410 participants were enrolled into the Open-Label Conversion and Titration Period and 281 participants were randomized into the Double-Blind Treatment Period, of which, 280 participants received study treatment.
Groups:
- Open ALO-02: Participants received AL0-02 extended-release capsules, orally (PO), twice daily (BID), at total daily doses of oxycodone from 20 to 160 milligrams (mg) in the Open-Label Conversion and Titration Period for 4 to 6 weeks; titration was at the discretion of the investigator.
- ALO-02 To Placebo: Participants received AL0-02 extended-release capsules PO BID at total daily doses of oxycodone from 20 to 160 mg in the Open-Label Conversion and Titration Period for 4 to 6 weeks; titration was at the discretion of the investigator. If a participant met protocol-defined treatment response criteria at the end of open-label Week 4, 5, or 6, the participant was randomized into the Double-Blind Treatment Period, underwent a double-blind gradual taper of ALO-02 to discontinue use over the first 2 weeks, and then received double-blind placebo capsules PO BID for 10 weeks.
- ALO-02 To ALO-02: Participants received AL0-02 extended-release capsules PO BID at total daily doses of oxycodone from 20 to 160 mg in the Open-Label Conversion and Titration Period for 4 to 6 weeks; titration was at the discretion of the investigator. If a participant met protocol-defined treatment response criteria at the end of open-label Week 4, 5, or 6, the participant was randomized into the Double-Blind Treatment Period, received a dummy-taper but continued to receive double-blind ALO-02 capsules PO BID at a fixed dose (specifically the ALO-02 fixed dose that had not changed with the 7 consecutive days prior to randomization) for 12 weeks.
Period: Open-Label Conversion + Titration Period
Arm/Group | Open ALO-02 | ALO-02 To Placebo | ALO-02 To ALO-02
Started | 410 | 0 (This phase commenced after the Open-Label Period.) | 0 (This phase commenced after the Open-Label Period.)
Completed | 281 | 0 (This phase commenced after the Open-Label Period.) | 0 (This phase commenced after the Open-Label Period.)
Not Completed | 129 | 0 | 0
Not completed — Withdrawal by Subject | 11 | 0 | 0
Not completed — Protocol Violation | 7 | 0 | 0
Not completed — Adverse Event | 57 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Not completed — Does not meet entrance criteria | 41 | 0 | 0
Not completed — Other - unspecified | 3 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Open ALO-02 | ALO-02 To Placebo | ALO-02 To ALO-02
Started | 0 (This phase preceded the Double-Blind Treatment Period.) | 134 | 146
Completed | 0 (This phase preceded the Double-Blind Treatment Period.) | 81 | 107
Not Completed | 0 | 53 | 39
Not completed — Withdrawal by Subject | 0 | 11 | 5
Not completed — Protocol Violation | 0 | 8 | 9
Not completed — Adverse Event | 0 | 9 | 14
Not completed — Lost to Follow-up | 0 | 3 | 6
Not completed — Insufficient clinical response | 0 | 16 | 4
Not completed — Other - unspecified | 0 | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Open ALO-02: Participants received AL0-02 extended-release capsules, orally PO BID at total daily doses of oxycodone from 20 to 160 mg in the Open-Label Conversion and Titration Period for 4 to 6 weeks; titration was at the discretion of the investigator.
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Age, Customized [Number; unit: Participants] — Age measure using NLM-defined categories.
  Participants
    Between 18 and 65 years | 364
    >=65 years | 46
Sex: Female, Male [Count of Participants; unit: Participants] — Gender
  Participants
    Female | 233
    Male | 177

OUTCOME MEASURES:

1. Primary Outcome: Change in Weekly Average Electronic Diary (eDiary) Numeric Rating Scale -Pain (NRS-Pain) Score From Randomization Baseline to Final 2 Weeks (Average of Weeks 11 and 12)
Description: Weekly average diary NRS-Pain scores were derived from the daily NRS-pain scale and calculated as the mean of the last 7 days. NRS-Pain scores based on an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain). Higher scores indicate greater pain.
Time Frame: Weeks 11 and 12
Population: Intent-to-Treat (ITT) Population: all participants who were randomized into the Double-Blind Treatment Period and received at least 1 dose of study drug after randomization; the averaged value for each participant from the 100 imputed datasets were used. Hybrid multiple and single imputation were applied, depending on reason for discontinuation.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 133 | 145
Units on a Scale | 1.23 (0.179) | 0.60 (0.168)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Null Hypothesis: No treatment difference. Power was 90%, 2-sided Alpha of 0.05, with assumed difference of 1 point and assumed standard deviation of 2.4 points; Test type: Superiority or Other; p = 0.0114, ANCOVA — No adjustment was made for multiple comparisons. Statistical significance was if unadjusted p was less than or equal to (<=) 0.05; Difference of LS Means = -0.62, 95% CI 2-sided [-1.11 to -0.14], Standard Error of Mean 0.246

2. Secondary Outcome: Change in Roland-Morris Disability Questionnaire (RMDQ) Total Score From Randomization Baseline to the End of Double-Blind Week 12 (or Final Visit).
Description: The RMDQ is a 24-item questionnaire designed to measure self-rated disability due to back pain. An individual participant's score can vary from 0 (no disability) to 24 (severe disability), with a lower score indicating better function; higher score indicating greater disability.
Time Frame: Week 12
Population: ITT Population; imputation using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 118 | 122
Units on a Scale | 0.50 (0.404) | 0.67 (0.393)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.7547, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and Baseline score and final total daily dose of Titration Period as covariates; Difference of LS Means = 0.18, 95% CI 2-sided [-0.94 to 1.29], Standard Error of Mean 0.565

3. Secondary Outcome: Percentage (%) of Participants With Shift in Patient Global Assessment (PGA) by Category With Baseline PGA Score of Very Good (1), Good (2), Fair (3), Poor (4), Very Poor (5) From Randomization Baseline to End of Double-Blind Week 12 (or Final Visit).
Description: Measure represents the score at Randomization Baseline / score at Week 12 (or Early Termination) in PGA, a global evaluation that utilizes a 5-point Likert scale with a score of 1 being the best (Very Good) and a score of 5 being the worst (Very Poor).
Time Frame: Randomization Baseline, Week 12
Population: ITT Population; percentage based on the number of participants who had non-missing values at Randomization Baseline and Week 12/early termination for each treatment. Imputation using LOCF method.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 130 | 137
Percentage of participants
  Very Good / Very Good | 5.4 | 11.7
  Very Good / Good | 6.2 | 2.9
  Very Good / Fair | 1.5 | 1.5
  Very Good / Poor | 0.8 | 0.0
  Very Good / Very Poor | 0.0 | 0.0
  Good / Very Good | 6.2 | 3.6
  Good / Good | 18.5 | 19.7
  Good / Fair | 4.6 | 6.6
  Good / Poor | 0.0 | 0.7
  Good / Very Poor | 0.0 | 0.0
  Fair / Very Good | 3.1 | 0.0
  Fair / Good | 17.7 | 21.2
  Fair / Fair | 23.1 | 26.3
  Fair / Poor | 0.8 | 2.2
  Fair / Very Poor | 0.0 | 0.0
  Poor / Very Good | 0.8 | 0.0
  Poor / Good | 2.3 | 1.5
  Poor / Fair | 4.6 | 2.2
  Poor / Poor | 1.5 | 0.0
  Poor / Very Poor | 0.0 | 0.0
  Very Poor / Very Good | 0.0 | 0.0
  Very Poor / Good | 1.5 | 0.0
  Very Poor / Fair | 1.5 | 0.0
  Very Poor / Poor | 0.0 | 0.0
  Very Poor / Very Poor | 0.0 | 0.0
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.1272, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) stratified by prior pain analgesic (opioid or non-opioid)

4. Secondary Outcome: Percentage of Participants With Improvement in Weekly Average eDiary NRS-Pain Scores From Screening to Final 2 Weeks of the Double-Blind Treatment Period (Average of Weeks 11 and 12) by Cumulative Percent Reduction of Greater or Equal to (≥) 20%
Description: Weekly average Diary NRS-pain scores are derived from the daily pain NRS and calculated as the mean of the last 7 days. Scores range from 0 equals (=) no pain to 10 = worst possible pain. Higher scores indicate greater pain.
Time Frame: Weeks 11 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
percentage of participants | 48.5 | 62.3
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0210, Cochran-Mantel-Haenszel; CMH was stratified by prior pain analgesic (opioid and non-opioid)

5. Secondary Outcome: Percentage of Participants With Improvement in Weekly Average eDiary NRS-Pain Scores From Screening to Final 2 Weeks of the Double-Blind Treatment Period (Average of Weeks 11 and 12) by Cumulative Percent Reduction ≥30%
Description: Weekly average Diary NRS-pain scores are derived from the daily pain NRS and calculated as the mean of the last 7 days. Scores range from 0 = no pain to 10 = worst possible pain. Higher scores indicate greater pain.
Time Frame: Weeks 11 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
percentage of participants | 44.0 | 57.5
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0248, Cochran-Mantel-Haenszel; The CMH test was stratified by prior pain analgesic (opioid or non-opioid)

6. Secondary Outcome: Percentage of Participants With Improvement in Weekly Average eDiary NRS-Pain Scores From Screening to Final 2 Weeks of the Double-Blind Treatment Period (Average of Weeks 11 and 12) by Cumulative Percent Reduction ≥40%
Description: as for outcome 5
Time Frame: Weeks 11 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
percentage of participants | 35.1 | 50.7
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0090, Cochran-Mantel-Haenszel; The CMH test was stratified by prior pain analgesic (opioid or non-opioid)

7. Secondary Outcome: Percentage of Participants With Improvement in Weekly Average eDiary NRS-Pain Scores From Screening to Final 2 Weeks of the Double-Blind Treatment Period (Average of Weeks 11 and 12) by Cumulative Percent Reduction ≥50%
Description: as for outcome 5
Time Frame: Weeks 11 and 12
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
percentage of participants | 29.9 | 39.7
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0874, Cochran-Mantel-Haenszel; The CMH test was stratified by prior pain analgesic (opioid or non-opioid)

8. Secondary Outcome: Change From Screening Period to End of Open-Label Treatment in Brief Pain Inventory - Short Form (BPI-sf): Worst Pain, Least Pain, Average Pain, Pain Right Now, Pain Severity Index, Pain Interference Index
Description: BPI-sf is an 11-item self-report questionnaire that is designed to assess the severity and impact of pain on daily functions. BPI-sf includes 4 questions that assess pain intensity (worst, least, average, right now) and 7 questions that assess impact of pain on daily functions (general activity, mood, walking ability, normal work, relations with other people, sleep, enjoyment of life). BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain. Pain Severity Index is the mean of the 4 pain scores (worst, least, average, and right now) on the BPI-sf; range is 0=No pain to 10=Pain as bad as you can imagine; A higher score indicates greater pain severity. Pain Interference Index is the mean of the scores for the 7 items of the BPI-sf; range is 0=Does not interfere to 10=Completely interferes.
Time Frame: Screening, Week 4, 5, or 6
Population: Titration Period Safety Population: defined as all participants who received any amount of ALO-02 capsules during the Open-Label Conversion and Titration Period; imputation using the LOCF method. n=number of participants contributing to the mean for the specified parameter.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Units on a Scale
  Worst Pain Score (n=400) | -3.3 (2.30)
  Least Pain Score (n=400) | -2.6 (2.33)
  Average Pain Score (n=400) | -3.0 (2.11)
  Pain Right Now (n=400) | -3.3 (2.41)
  Pain Severity Index (n=400) | -3.1 (2.07)
  Pain Interference Index (n=401) | -2.8 (2.32)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Worst Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Least Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Average Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Pain Right Now; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Pain Severity Index; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Open ALO-02; Change from Screening Period value to end of the OL Period for Pain Interference Index; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

9. Secondary Outcome: Change From Screening Period to Randomization Baseline in BPI-sf: Worst Pain, Least Pain, Average Pain, Pain Right Now, Pain Severity Index, Pain Interference Index
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain. Pain Severity Index is the mean of the 4 pain scores (worst, least, average, and right now) on the BPI-sf; range is 0=No pain to 10=Pain as bad as you can imagine; A higher score indicates greater pain severity. Pain Interference Index is the mean of the scores for the 7 items of the BPI-sf; range is 0=Does not interfere to 10=Completely interferes.
Time Frame: Screening, Randomization Baseline
Population: ITT Population - observed cases; n=number of participants assessed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 279
units on scale
  Worst Pain Score (n=279) | -4.2 (1.83)
  Least Pain Score (n=279) | -3.4 (2.04)
  Average Pain Score (n=279) | -3.8 (1.60)
  Pain Right Now (n=279) | -4.2 (1.95)
  Pain Severity Index (n=279) | -3.9 (1.63)
  Pain Interference Index (n=279) | -3.4 (2.16)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Worst Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Least Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Average Pain Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Pain Right Now; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Pain Severity Index; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Pain Interference Index; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

10. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Worst Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for worst pain at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,135) | 1.00 (0.160) | 0.38 (0.155)
  Week 4 (n=111,125) | 1.15 (0.179) | 0.51 (0.168)
  Week 8 (n=89,113) | 0.86 (0.205) | 0.49 (0.180)
  Week 12/Early Termination (ET)(n=131,138) | 1.45 (0.176) | 0.47 (0.170)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0056, ANCOVA; Difference of LS Means = -0.62, 95% CI 2-sided [-1.06 to -0.18], Standard Error of Mean 0.222 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Randomization Baseline score and final total daily dose of the Titration Period as covariates
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p = 0.0090, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-1.12 to -0.16], Standard Error of Mean 0.243 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.1684, ANCOVA; Difference of LS Means = -0.37, 95% CI 2-sided [-0.91 to 0.16], Standard Error of Mean 0.271 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.98, 95% CI 2-sided [-1.46 to -0.50], Standard Error of Mean 0.244 — [estimate comment as in outcome 10, analysis 1]

11. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Least Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation by LOCF; n=number of participants assessed for least pain at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,135) | 0.74 (0.139) | 0.34 (0.134)
  Week 4 (n=111,125) | 0.94 (0.147) | 0.06 (0.138)
  Week 8 (n=89,112) | 0.83 (0.171) | 0.19 (0.151)
  Week 12/ET(n=131,138) | 1.13 (0.151) | 0.28 (0.147)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0412, ANCOVA; Difference of LS Means = -0.40, 95% CI 2-sided [-0.78 to -0.02], Standard Error of Mean 0.193 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.87, 95% CI 2-sided [-1.27 to -0.48], Standard Error of Mean 0.201 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.0055, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-1.08 to -0.19], Standard Error of Mean 0.226 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.86, 95% CI 2-sided [-1.27 to -0.44], Standard Error of Mean 0.210 — [estimate comment as in outcome 10, analysis 1]

12. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Average Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for average pain at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=125,135) | 1.01 (0.137) | 0.36 (0.132)
  Week 4 (n=111,124) | 1.04 (0.156) | 0.30 (0.147)
  Week 8 (n=88,112) | 0.99 (0.179) | 0.35 (0.157)
  Week 12/ET (n=131,138) | 1.27 (0.159) | 0.39 (0.154)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0007, ANCOVA; Difference of LS Means = -0.65, 95% CI 2-sided [-1.02 to -0.27], Standard Error of Mean 0.190 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p = 0.0006, ANCOVA; Difference of LS Means = -0.74, 95% CI 2-sided [-1.16 to -0.32], Standard Error of Mean 0.213 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.0070, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-1.11 to -0.18], Standard Error of Mean 0.236 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.88, 95% CI 2-sided [-1.31 to -0.44], Standard Error of Mean 0.221 — [estimate comment as in outcome 10, analysis 1]

13. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Right Now
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for pain right now at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,135) | 1.04 (0.149) | 0.40 (0.144)
  Week 4 (n=111,125) | 1.03 (0.157) | 0.24 (0.148)
  Week 8 (n=88,112) | 1.04 (0.200) | 0.33 (0.176)
  Week 12/ET (n=131,138) | 1.43 (0.166) | 0.36 (0.161)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0022, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-1.05 to -0.23], Standard Error of Mean 0.207 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p = 0.0003, ANCOVA; Difference of LS Means = -0.79, 95% CI 2-sided [-1.21 to -0.37], Standard Error of Mean 0.214 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.0078, ANCOVA; Difference of LS Means = -0.71, 95% CI 2-sided [-1.23 to -0.19], Standard Error of Mean 0.264 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -1.07, 95% CI 2-sided [-1.52 to -0.62], Standard Error of Mean 0.231 — [estimate comment as in outcome 10, analysis 1]

14. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Severity Index
Description: Pain Severity Index is the mean of the 4 pain scores (worst, least, average, and right now) on the BPI-sf; range is 0=No pain to 10=Pain as bad as you can imagine; a higher score indicates greater pain severity.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for pain severity index at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=125,135) | 0.95 (0.136) | 0.37 (0.131)
  Week 4 (n=111,124) | 1.04 (0.145) | 0.28 (0.137)
  Week 8 (n=88,112) | 0.95 (0.173) | 0.34 (0.152)
  Week 12/ET (n=131,138) | 1.32 (0.149) | 0.38 (0.144)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0022, ANCOVA; Difference of LS Means = -0.58, 95% CI 2-sided [-0.95 to -0.21], Standard Error of Mean 0.189 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference of LS Means = -0.76, 95% CI 2-sided [-1.15 to -0.37], Standard Error of Mean 0.198 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.0078, ANCOVA; Difference of LS Means = -0.61, 95% CI 2-sided [-1.06 to -0.16], Standard Error of Mean 0.228 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.95, 95% CI 2-sided [-1.35 to -0.54], Standard Error of Mean 0.207 — [estimate comment as in outcome 10, analysis 1]

15. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Interference Index
Description: Pain Interference Index is the mean of the scores for the 7 items of the BPI-sf; range is 0=Does not interfere to 10=Completely interferes.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for pain interference index at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,135) | 0.77 (0.135) | 0.36 (0.130)
  Week 4 (n=111,127) | 0.92 (0.139) | 0.43 (0.129)
  Week 8 (n=89,113) | 0.64 (0.168) | 0.47 (0.148)
  Week 12/ET (n=131,138) | 1.14 (0.149) | 0.49 (0.145)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 2; Test type: Superiority or Other; p = 0.0285, ANCOVA; Difference of LS Means = -0.41, 95% CI 2-sided [-0.78 to -0.04], Standard Error of Mean 0.188 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 4; Test type: Superiority or Other; p = 0.0106, ANCOVA; Difference of LS Means = -0.48, 95% CI 2-sided [-0.85 to -0.11], Standard Error of Mean 0.188 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 8; Test type: Superiority or Other; p = 0.4529, ANCOVA; Difference of LS Means = -0.17, 95% CI 2-sided [-0.60 to 0.27], Standard Error of Mean 0.222 — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline to Week 12/Early Termination; Test type: Superiority or Other; p = 0.0018, ANCOVA; Difference of LS Means = -0.65, 95% CI 2-sided [-1.06 to -0.25], Standard Error of Mean 0.207 — [estimate comment as in outcome 10, analysis 1]

16. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Worst Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8 and 12
Population: as for outcome 10
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,134) | -3.09 (0.186) | -3.80 (0.181)
  Week 4 (n=111,124) | -3.01 (0.203) | -3.74 (0.192)
  Week 8 (n=89,112) | -3.16 (0.238) | -3.72 (0.212)
  Week 12/ET (n=131,137) | -2.63 (0.207) | -3.73 (0.203)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0061, ANCOVA; Difference of LS Means = -0.71, 95% CI 2-sided [-1.22 to -0.20], Standard Error of Mean 0.258 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0087, ANCOVA; Difference of LS Means = -0.73, 95% CI 2-sided [-1.28 to -0.19], Standard Error of Mean 0.277 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.0769, ANCOVA; Difference of LS Means = -0.56, 95% CI 2-sided [-1.18 to 0.06], Standard Error of Mean 0.315 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/Early Termination; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference of LS Means = -1.10, 95% CI 2-sided [-1.67 to -0.53], Standard Error of Mean 0.289 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

17. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Least Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; Higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: ITT Population - imputed values at early termination. Imputation using the LOCF method; n=number of participants assessed for least pain at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,134) | -2.55 (0.162) | -3.05 (0.157)
  Week 4 (n=111,124) | -2.40 (0.171) | -3.29 (0.162)
  Week 8 (n=89,111) | -2.44 (0.199) | -3.21 (0.178)
  Week 12/ET (n=131,137) | -2.14 (0.175) | -3.12 (0.171)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0250, ANCOVA; Difference of LS Means = -0.51, 95% CI 2-sided [-0.95 to -0.06], Standard Error of Mean 0.224 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference of LS Means = -0.89, 95% CI 2-sided [-1.36 to -0.43], Standard Error of Mean 0.234 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.0038, ANCOVA; Difference of LS Means = -0.77, 95% CI 2-sided [-1.29 to -0.25], Standard Error of Mean 0.263 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -0.98, 95% CI 2-sided [-1.46 to -0.50], Standard Error of Mean 0.243 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

18. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Average Pain
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=125,134) | -2.63 (0.154) | -3.43 (0.150)
  Week 4 (n=111,123) | -2.76 (0.172) | -3.55 (0.164)
  Week 8 (n=88,111) | -2.71 (0.205) | -3.50 (0.182)
  Week 12/ET (n=131,137) | -2.39 (0.176) | -3.43 (0.172)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0002, ANCOVA; Difference of LS Means = -0.80, 95% CI 2-sided [-1.22 to -0.38], Standard Error of Mean 0.214 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0010, ANCOVA; Difference of LS Means = -0.78, 95% CI 2-sided [-1.25 to -0.32], Standard Error of Mean 0.235 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.0041, ANCOVA; Difference of LS Means = -0.79, 95% CI 2-sided [-1.32 to -0.25], Standard Error of Mean 0.271 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -1.04, 95% CI 2-sided [-1.52 to -0.56], Standard Error of Mean 0.245 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

19. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Right Now
Description: BPI-sf scores range from 0=No pain to 10=Pain as bad as you can imagine; higher scores indicate greater pain.
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 13
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,134) | -3.12 (0.170) | -3.72 (0.165)
  Week 4 (n=111,124) | -3.15 (0.187) | -3.82 (0.177)
  Week 8 (n=88,111) | -3.00 (0.232) | -3.71 (0.206)
  Week 12/ET (n=131,137) | -2.72 (0.189) | -3.74 (0.186)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0115, ANCOVA; Difference of LS Means = -0.60, 95% CI 2-sided [-1.06 to -0.14], Standard Error of Mean 0.236 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0099, ANCOVA; Difference of LS Means = -0.66, 95% CI 2-sided [-1.17 to -0.16], Standard Error of Mean 0.256 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.0222, ANCOVA; Difference of LS Means = -0.71, 95% CI 2-sided [-1.31 to -0.10], Standard Error of Mean 0.307 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/ Early Termination; Test type: Superiority or Other; p = 0.0001, ANCOVA; Difference of LS Means = -1.02, 95% CI 2-sided [-1.54 to -0.50], Standard Error of Mean 0.264 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

20. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Severity Index
Description: as for outcome 14
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=125,134) | -2.83 (0.157) | -3.50 (0.152)
  Week 4 (n=111,123) | -2.83 (0.172) | -3.60 (0.164)
  Week 8 (n=88,111) | -2.80 (0.205) | -3.53 (0.182)
  Week 12/ET (n=131,137) | -2.47 (0.174) | -3.51 (0.171)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0025, ANCOVA; Difference of LS Means = -0.66, 95% CI 2-sided [-1.09 to -0.24], Standard Error of Mean 0.218 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0012, ANCOVA; Difference of LS Means = -0.77, 95% CI 2-sided [-1.23 to -0.31], Standard Error of Mean 0.235 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.0078, ANCOVA; Difference of LS Means = -0.73, 95% CI 2-sided [-1.27 to -0.19], Standard Error of Mean 0.272 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/Early Termination; Test type: Superiority or Other; p < 0.0001, ANCOVA; Difference of LS Means = -1.04, 95% CI 2-sided [-1.52 to -0.56], Standard Error of Mean 0.243 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

21. Secondary Outcome: Change From Screening to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in BPI-sf Scores of Pain Interference Index
Description: as for outcome 15
Time Frame: Weeks 2, 4, 8, and 12
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a Scale
  Week 2 (n=126,134) | -2.58 (0.164) | -2.99 (0.160)
  Week 4 (n=111,126) | -2.52 (0.175) | -2.99 (0.164)
  Week 8 (n=89,112) | -2.72 (0.198) | -2.87 (0.176)
  Week 12/ET (n=131,137) | -2.24 (0.176) | -2.88 (0.172)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 2; Test type: Superiority or Other; p = 0.0727, ANCOVA; Difference of LS Means = -0.41, 95% CI 2-sided [-0.86 to 0.04], Standard Error of Mean 0.228 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 4; Test type: Superiority or Other; p = 0.0501, ANCOVA; Difference of LS Means = -0.47, 95% CI 2-sided [-0.94 to 0.00], Standard Error of Mean 0.238 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 8; Test type: Superiority or Other; p = 0.5704, ANCOVA; Difference of LS Means = -0.15, 95% CI 2-sided [-0.67 to 0.37], Standard Error of Mean 0.262 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening to Week 12/ Early Termination; Test type: Superiority or Other; p = 0.0096, ANCOVA; Difference of LS Means = -0.64, 95% CI 2-sided [-1.12 to -0.16], Standard Error of Mean 0.245 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate

22. Secondary Outcome: Area Under the Curve (AUC) of eDiary NRS-Pain Scores From Randomization Baseline to Final 2 Weeks of the Double-Blind Treatment Period (Weeks 11 and 12)
Description: NRS-Pain scores based on an 11-point numerical rating scale from 0 (no pain) to 10 (worst possible pain). AUC was calculated using daily change from Baseline scores from Baseline until the last dose date in the Double-Blind Treatment Period. AUC was calculated for each participant using the linear trapezoidal method. Higher scores indicate greater pain.
Time Frame: Randomization Baseline, Weeks 11 and 12
Population: ITT Population; linear interpolation was used for internal missing values, with addition of 0 to the AUC for missing values from early discontinuation.
Measure: Least Squares Mean (Standard Error); unit: Change in units on a scale*days
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Change in units on a scale*days | 39.00 (7.914) | 11.25 (7.636)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0120, ANCOVA; Difference of LS Means = -27.75, 95% CI 2-sided [-49.34 to -6.16], Standard Error of Mean 10.968 — Difference between treatment groups evaluated by ANCOVA with treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Randomization Baseline score and final total daily dose of the Titration Period as covariates

23. Secondary Outcome: Average Daily Use of Rescue Acetaminophen (Milligrams Per Day [mg/Day]) During the Double-Blind Treatment Period
Description: The amount of acetaminophen administered for each treatment during the Double-Blind Treatment Period. Average daily use calculated as: total dose of rescue medication during Double-Blind Period divided by the number of days in Double-Blind Period.
Time Frame: Daily from Day 1 of the Double-Blind Period through Week 12
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: Average mg/day
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Average mg/day | 207.84 (36.436) | 203.97 (34.851)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.9390, ANCOVA; Difference of LS Means = -3.87, 95% CI 2-sided [-103.29 to 95.55], Standard Error of Mean 50.500 — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the average daily rescue acetaminophen during the Titration Period and final total daily study medication dose of the Titration Period as covariates

24. Secondary Outcome: Percentage of Participants With a 20%, 30%, 40%, or 50% Analgesic Response From Screening Period to End of Open-Label Treatment
Description: The percentage of analgesic response is defined as: (rolling 7-day mean pain score during Titration Period - Screening Period pain intensity score) divided by Screening Period pain intensity score times100.
Time Frame: Screening, Week 4, 5 or 6
Population: Titration Period Safety Population; an event was defined as a participant with 20%, 30%, 40%, or 50% analgesic response from Screening.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 398
Percentage of participants
  Participants with 20% Analgesic Response | 85.2
  Participants with 30% Analgesic Response | 78.9
  Participants with 40% Analgesic Response | 67.3
  Participants with 50% Analgesic Response | 49.7

25. Secondary Outcome: Median Time to 20%, 30%, 40%, or 50% Analgesic Response From Screening Period to End of Open-Label Treatment
Description: The percentage of analgesic response is defined as: (rolling 7-day mean pain score during Titration Period minus (-) Screening Period pain intensity score) divided by Screening Period pain intensity score times 100. An event was defined as a participant with 20, 30, 40, or 50% analgesic response from Screening. If there was no event for a participant, time to the event was considered censored at Day 42 of the Titration Period or before Day 42 of the Titration Period at the time of the last diary pain score. The survival duration begins on the date of first dose of study drug in the Titration Period and is calculated as the [date of event or last diary pain score - date of first dose in Titration Period +1].
Time Frame: Screening, Week 4, 5, or 6
Population: as for outcome 24
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 398
days
  Time to 20% Analgesic Response from Screening | 15 [14.0 to 17.0]
  Time to 30% Analgesic Response from Screening | 21 [19.0 to 23.0]
  Time to 40% Analgesic Response from Screening | 28 [26.0 to 30.0]
  Time to 50% Analgesic Response from Screening | 35 [32.0 to 38.0]

26. Secondary Outcome: Percentage of Participants With a 20%, 30%, 40%, or 50% Analgesic Response From Screening Period to Randomization Baseline
Description: The percentage of analgesic response is defined as: (rolling 7-day mean pain score during Titration Period - Screening Period pain intensity score) divided by Screening Period pain intensity score times 100.
Time Frame: Screening, Randomization Baseline (up to 6 weeks)
Population: ITT Population; an event was defined as a participant with 20%, 30%, 40%, or 50% analgesic response from Screening.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 278
Percentage of participants
  Participants with 20% Analgesic Response | 99.3
  Participants with 30% Analgesic Response | 95.3
  Participants with 40% Analgesic Response | 86.0
  Participants with 50% Analgesic Response | 64.0

27. Secondary Outcome: Median Time to 20%, 30%, 40%, or 50% Analgesic Response From Screening Period to Randomization Baseline
Description: The percentage of analgesic response is defined as: (rolling 7-day mean pain score during Titration Period - Screening Period pain intensity score) divided by Screening Period pain intensity score times 100. If there was no event for a participant, time to the event was considered censored at Day 42 of the Titration Period or before Day 42 of the Titration Period at the time of the last diary pain score. The survival duration begins on the date of first dose of study drug in the Titration Period and is calculated as the [date of event or last diary pain score - date of first dose in Titration Period +1].
Time Frame: Screening, Randomization Baseline (up to 6 weeks)
Population: ITT Population; an event was defined as a participant with 20%, 30%, 40% or 50% analgesic response from Screening.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 278
days
  Time to 20% Analgesic Response | 14 [13.0 to 16.0]
  Time to 30% Analgesic Response | 20 [17.0 to 22.0]
  Time to 40% Analgesic Response | 26 [23.0 to 28.0]
  Time to 50% Analgesic Response | 33 [30.0 to 35.0]

28. Secondary Outcome: Percentage of Participants With a 20%, 30%, 40%, or 50% Loss of Analgesic Response From Randomization Baseline During the Double-Blind Treatment Period
Description: The percentage of lost analgesic response is defined as: (rolling 7-day mean pain score during Double-Blind Period - Randomization Baseline pain intensity score) divided by Randomization Baseline pain intensity score times 100. If there was no event for a participant, time to the event was considered censored at Day 84 or before Day 84 at the time of the last diary pain score. The survival duration began on the date of first dose of study drug in the Double-Blind Period and was calculated as the [date of event or last diary pain score - date of first dose in Double-Blind Treatment +1].
Time Frame: Randomization Baseline, up to Week 12
Population: ITT Population; an event was defined as a participant with 20%, 30%, 40%, or 50% loss of analgesic response from Randomization Baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 132 | 143
Percentage of participants
  Participants with 20% Loss of Analgesic Response | 72.0 | 54.5
  Participants with 30% Loss of Analgesic Response | 64.4 | 46.2
  Participants with 40% Loss of Analgesic Response | 57.6 | 34.3
  Participants with 50% Loss of Analgesic Response | 50.8 | 31.5

29. Secondary Outcome: Median Time to 20%, 30%, 40%, or 50% Loss of Analgesic Response From Baseline During the Double-Blind Treatment Period
Description: The percentage of lost analgesic response was defined as: (rolling seven day mean pain score during Double-Blind Period - Randomization Baseline pain intensity score) divided by Randomization Baseline pain intensity score times 100. If there was no event for a participant, time to the event was considered censored at Day 84 or before Day 84 at the time of the last diary pain score. The survival duration began on the date of first dose of study drug in the Double-Blind Period and was calculated as the [date of event or last diary pain score - date of first dose in Double-Blind Treatment +1].
Time Frame: Randomization Baseline, up to Week 12
Population: as for outcome 28
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 132 | 143
days
  Time to 20% Loss of Analgesic Response | 12 [8.0 to 17.0] | 31 [18.0 to NA] — Number of participants with loss of response was too low to estimate the 95% confidence interval upper limit.
  Time to 30% Loss of Analgesic Response | 21 [15.0 to 39.0] | NA [32.0 to NA] — Number of participants with loss of response was too low to estimate the median time and 95% confidence interval upper limit.
  Time to 40% Loss of Analgesic Response | 41 [21.0 to 61.0] | NA [NA to NA] — Number of participants with loss of response was too low to estimate the median time and 95% confidence interval upper and lower limits.
  Time to 50% Loss of Analgesic Response | 62 [24.0 to NA] — Number of participants with loss of response was too low to estimate the 95% confidence interval upper limit. | NA [NA to NA] — Number of participants with loss of response was too low to estimate the median time and 95% confidence interval upper and lower limits.
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Time to 20% loss of analgesic response; Test type: Superiority or Other; p = 0.0014, Wilcoxon test, survival analysis; P-value from Wilcoxon test with treatment and opioid stratum as factors
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Time to 30% loss of analgesic response; Test type: Superiority or Other; p = 0.0024, Wilcoxon test, survival analysis; P-value from Wilcoxon test with treatment and opioid stratum as factors
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Time to 40% loss of analgesic response; Test type: Superiority or Other; p = 0.0006, Wilcoxon test, survival analysis; P-value from Wilcoxon test with treatment and opioid stratum as factors
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Time to 50% loss of analgesic response; Test type: Superiority or Other; p = 0.0021, Wilcoxon test, survival analysis; P-value from Wilcoxon test with treatment and opioid stratum as factors

30. Secondary Outcome: Percentage of Participants Discontinuing Treatment for Investigator-Reported Lack of Efficacy
Description: If there was no event for a participant, time to the event was considered censored at Day 84 or before Day 84 at time of treatment discontinuation for another reason.
Time Frame: Week 1 up to Week 12
Population: ITT Population; an event was defined as a participant with treatment discontinuation for investigator-reported lack of efficacy.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Percentage of participants | 11.9 | 2.7

31. Secondary Outcome: Median Time to Treatment Discontinuation for Investigator-Reported Lack of Efficacy During the Double-Blind Treatment Period
Description: If there was no event for a participant, time to the event was considered censored at Day 84 or before Day 84 at time of treatment discontinuation for another reason. The survival duration begins on the date of first dose in the Double-Blind period and is calculated as the [date of event or discontinuation - date of first dose in Double-Blind Period +1].
Time Frame: Week 1 up to Week 12
Population: as for outcome 30
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
days | NA [NA to NA] — Incidence of discontinuation from investigator-reported lack of efficacy was too low to estimate median. | NA [NA to NA] — Incidence of discontinuation from investigator-reported lack of efficacy was too low to estimate median.
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.006, Wilcoxon test, survival analysis; P-value from Wilcoxon test with treatment and opioid stratum as factors

32. Secondary Outcome: Clinical Opiate Withdrawal Scale (COWS) Total Score During the Open-Label Titration Period
Description: The COWS contains 11 common opiate withdrawal signs or symptoms rated by the investigator or designee who, for each item, checked the number that best described the participant's signs or symptoms. The minimum total COWS score is 0, the maximum is 48. Higher scores indicate a worse outcome. The summed score of the 11 items was used to assess a participant's level of opiate withdrawal.
Time Frame: Screening, Weeks 1, 2, 3, 4, 5, and 6
Population: Titration Period Safety Population. Only participants with values at both Screening and each respective visit were included in the change from screening analysis; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Units on a scale
  Screening (n=387) | 0.6 (1.09)
  Week 1 (n=353) | 0.6 (1.04)
  Change from Screening at Week 1 (n=333) | 0.0 (1.20)
  Week 2 (n=327) | 0.5 (1.08)
  Change from Screening at Week 2 (n=308) | 0.0 (1.25)
  Week 3 (n=316) | 0.5 (0.92)
  Change from Screening at Week 3 (n=295) | -0.1 (1.21)
  Week 4 (n=210) | 0.6 (0.94)
  Change from Screening at Week 4 (n=194) | 0.0 (1.27)
  Week 5 (n=138) | 0.6 (0.82)
  Change from Screening at Week 5 (n=131) | -0.1 (1.15)
  Week 6/ET (n=375) | 0.6 (0.99)
  Change from Screening at Week 6 (n=352) | 0.0 (1.28)
  Maximum Titration Period (MTP) Value (n=375) | 1.2 (1.42)
  Change from screening to MTP Value (n=352) | 0.6 (1.54)

33. Secondary Outcome: COWS Total Score During the Double-Blind Treatment Period
Description: as for outcome 32
Time Frame: Randomization Baseline, Weeks 1, 2, 4, 8, and 12
Population: Double-Blind Safety Population. Only participants with values at both Randomization Baseline and each respective visit were included in the change from Randomization Baseline analysis; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a scale
  Randomization Baseline (n=134,146) | 0.6 (0.85) | 0.4 (0.73)
  Week 1 (n=111,133) | 0.8 (1.62) | 0.6 (1.13)
  Change from Baseline at Week 1 (n=111,133) | 0.3 (1.69) | 0.3 (1.12)
  Week 2 (n=115,128) | 0.8 (1.28) | 0.7 (1.19)
  Change from Baseline at Week 2 (n=115,128) | 0.2 (1.45) | 0.3 (1.10)
  Week 4 (n=106,123) | 0.6 (0.90) | 0.4 (0.66)
  Change from Baseline at Week 4 (n=106,123) | 0.1 (1.10) | 0.1 (0.79)
  Week 8 (n=87,107) | 0.6 (1.02) | 0.6 (1.10)
  Change from Baseline at Week 8 (n=87,107) | 0.1 (1.03) | 0.2 (1.06)
  Week 12/ET (n=126,140) | 0.7 (1.55) | 0.6 (1.17)
  Change from Baseline at Week 12/ET(n=126,140) | 0.2 (1.61) | 0.2 (1.21)
  Max. Double-Blind Period (DBP) Value (n=126,140) | 1.4 (1.84) | 1.3 (1.60)
  Change from Baseline to max. DBP Value (n=126,140) | 0.9 (1.90) | 0.9 (1.53)

34. Secondary Outcome: COWS Total Score During the Post-Treatment Period
Description: as for outcome 32
Time Frame: Follow-Up (FU) Weeks 1 and 2
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 94 | 108
Units on a scale
  FU Week 1 (n=68,83) | 0.6 (0.72) | 0.6 (0.91)
  Change from Baseline at FU Week 1 (n=68,83) | 0.1 (0.90) | 0.2 (0.99)
  FU Week 2 (n=78,91) | 0.5 (0.70) | 0.9 (1.74)
  Change from Baseline at FU Week 2 (n=78,91) | -0.1 (1.12) | 0.7 (1.83)
  Max.FU Period Value (n=94,108) | 0.7 (0.76) | 1.1 (1.67)
  Change to max. FU Period Value (n=94,108) | 0.1 (1.08) | 0.7 (1.74)

35. Secondary Outcome: Percentage of Participants With Opiate Withdrawal During the Open-Label Titration Period by COWS Category
Description: The COWS contains 11 common opiate withdrawal signs or symptoms rated by the investigator or designee who, for each item, checked the number that best described the participant's signs or symptoms. The minimum total COWS score is 0, the maximum is 48. The summed score of the 11 items was used to assess a participant's level of opiate withdrawal. The scores are assessed as follows: 5-12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal.
Time Frame: Screening, Weeks 1, 2, 3, 4, 5, 6 (or Early Termination)
Population: Titration Period Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Percentage of participants
  Screening COWS less than(<)5 (n=387) | 98.4
  Screening COWS=5-12 (n=387) | 1.6
  Week 1 COWS <5 (n=353) | 99.2
  Week 1 COWS=5-12 (n=353) | 0.8
  Week 2 COWS <5 (n=327) | 98.8
  Week 2 COWS 5-12 (n=327) | 1.2
  Week 3 COWS <5 (n=316) | 99.1
  Week 3 COWS 5-12 (n=316) | 0.9
  Week 4 COWS <5 (n=210) | 99.5
  Week 4 COWS 5-12 (n=210) | 0.5
  Week 5 COWS <5 (n=138) | 100
  Week 6 COWS <5 (n=375) | 98.9
  Week 6 COWS 5-12 (n=375) | 1.1
  Max. Titration Period Value COWS <5 (n=375) | 96.8
  Max. Titration Period Value COWS 5-12 (n=375) | 3.2

36. Secondary Outcome: Percentage of Participants With Opiate Withdrawal During the Double-Blind Treatment Period by COWS Category
Description: as for outcome 35
Time Frame: Randomization Baseline, Weeks 1, 2, 4, 8, 12 (or Early Termination)
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Percentage of participants
  Randomization Baseline COWS <5 (n=134,146) | 100 | 100
  Week 1 COWS <5 (n=111,133) | 99.1 | 98.5
  Week 1 COWS 5-12 (n=111,133) | 0 | 1.5
  Week 1 COWS 13-24 (n=111,133) | 0.9 | 0
  Week 2 COWS <5 (n=115,128) | 99.1 | 98.4
  Week 2 COWS 5-12 (n=115,128) | 0.9 | 1.6
  Week 4 COWS <5 (n=106,123) | 99.1 | 100
  Week 4 COWS 5-12 (n=106,123) | 0.9 | 0
  Week 8 COWS <5 (n=87,107) | 100 | 98.1
  Week 8 COWS 5-12 (n=87,107) | 0 | 1.9
  Week 12/ET COWS <5 (n=126,140) | 98.4 | 97.9
  Week 12/ET COWS 5-12 (n=126,140) | 0.8 | 2.1
  Week 12/ET COWS 13-24 (n=126,140) | 0.8 | 0
  Max. DBP Value COWS <5 (n=126,140) | 97.6 | 95.0
  Max. DBP Value COWS 5-12 (n=126,140) | 1.6 | 5.0
  Max. DBP Value COWS 13-24 (n=126,140) | 0.8 | 0

37. Secondary Outcome: Percentage of Participants With Opiate Withdrawal During Post-Treatment by COWS Category
Description: as for outcome 35
Time Frame: Follow-Up Weeks 1 and 2
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 94 | 108
Percentage of participants
  FU Week 1 COWS <5 (n=68,83) | 100.0 | 100.0
  FU Week 2 COWS <5 (n=78,91) | 100 | 95.6
  FU Week 2 COWS=5-12 (n=78,91) | 0 | 4.4
  Maximum FU Period COWS <5 (n=94,108) | 100.0 | 96.3
  Maximum FU Period COWS=5-12 (n=94,108) | 0 | 3.7

38. Secondary Outcome: Subjective Opiate Withdrawal Scale (SOWS) During the Open-Label Titration Period
Description: The SOWS was completed daily by the participant during any of the 2-week tapers from study drug, as well as at each study visit, using an eDiary device, and contains 16 symptoms of opiate withdrawal rated by the participant (Scale of 0 to 4: 0 = not at all, 1 = a little, 2= moderately, 3= quite a bit, 4 = extremely). The sum of the scores on each item was the total SOWS score; the minimum possible SOWS score was 0, the maximum 64. Higher scores indicate a worse outcome.
Time Frame: Screening, Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Units on a scale
  Screening (n=395) | 4.1 (4.92)
  Week 1 (n=355) | 3.5 (4.31)
  Change from Screening at Week 1 (n=346) | -0.7 (4.71)
  Week 2 (n=329) | 3.0 (3.66)
  Change from Screening at Week 2 (n=320) | -1.2 (4.64)
  Week 3 (n=311) | 2.7 (4.17)
  Change from Screening at Week 3 (n=304) | -1.4 (5.24)
  Week 4 (n=206) | 2.2 (2.92)
  Change from Screening at Week 4 (n=199) | -2.1 (4.92)
  Week 5 (n=139) | 2.2 (2.96)
  Change from Screening at Week 5 (n=133) | -2.4 (4.42)
  Week 6/ET (n=369) | 3.0 (4.41)
  Change from Screening at Week 6/ET (n=359) | -1.2 (5.36)
  Max. SOWS (Titration Period) (n=369) | 4.9 (5.35)
  Change from Screening at Max. SOWS (n=359) | 0.7 (5.51)

39. Secondary Outcome: SOWS Total Score During the Double-Blind Treatment Period
Description: as for outcome 38
Time Frame: Randomization Baseline, Weeks 1, 2, 4, 8, and 12
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a scale
  Randomization Baseline (n=134,146) | 2.4 (3.88) | 1.5 (2.20)
  Week 1 (n=134,143) | 3.0 (4.27) | 2.3 (3.69)
  Change from Baseline at Week 1 (n=134,143) | 0.6 (4.08) | 0.8 (2.93)
  Week 2 (n=123,135) | 3.5 (6.56) | 1.9 (3.11)
  Change from Baseline at Week 2 (n=123,135) | 1.1 (5.37) | 0.3 (2.64)
  Max. SOWS, First 2 Weeks of Period (n=134,143) | 6.3 (7.72) | 4.4 (5.11)
  Week 4 (n=105,122) | 2.5 (3.91) | 2.1 (3.42)
  Change from Baseline at Week 4 (n=105,122) | 0.1 (3.57) | 0.5 (2.39)
  Week 8 (n=85,110) | 2.4 (4.48) | 2.1 (3.37)
  Change from Baseline at Week 8 (n=85,110) | 0.1 (3.83) | 0.6 (2.92)
  Week 12 (n=134,143) | 3.3 (5.70) | 2.4 (3.85)
  Change from Baseline at Week 12 (n=134,143) | 0.9 (5.11) | 0.9 (3.01)
  Max. SOWS (Double-Blind Period) (n=134,143) | 6.7 (7.77) | 5.2 (5.89)
  Change from Baseline at max. SOWs (n=134,143) | 4.3 (5.82) | 3.7 (5.14)

40. Secondary Outcome: SOWS Total Score During the Post-Treatment Period
Description: as for outcome 38
Time Frame: Follow-Up Weeks 1 and 2
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 96 | 110
Units on a scale
  FU Week 1 (n=94,108) | 2.6 (4.91) | 2.3 (3.69)
  Change from Baseline at FU Week 1 (n=94,108) | 0.2 (4.12) | 0.8 (3.21)
  FU Week 2 (n=95,109) | 2.7 (5.26) | 2.5 (3.67)
  Change from Baseline at FU Week 2 (n=95,109) | 0.2 (4.49) | 1.0 (3.35)
  Max. SOWS (FU Period)(n=96,110) | 4.7 (6.73) | 4.5 (5.45)
  Change from Baseline at Max. SOWS, (n=96,110) | 2.2 (5.31) | 3.0 (4.77)

41. Secondary Outcome: Change From Screening Period to End of Open-Label Titration Period in Roland-Morris Disability Questionnaire (RMDQ) Total Score for All Participants
Description: RMDQ is a 24-item questionnaire designed to measure self-rated disability due to back pain the same day the questionnaire is completed. An individual participant's score could have ranged from 0 (no disability) to 24 (severe disability), with a lower score indicating better function; higher scores indicating greater disability.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Units on a scale
  Screening (n=405) | 12.7 (5.42)
  End of Open-Label Titration Period (n=345) | 9.0 (5.62)
  Change from Screening (n=343) | -3.9 (4.91)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to the End of Open-Label Titration Period; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

42. Secondary Outcome: Change From Screening Period to Randomization Baseline in RMDQ Total Score
Description: RMDQ is a 24-item questionnaire designed to measure self-rated disability due to back pain the same day the questionnaire is completed. An individual participant's score could have ranged from 0 (no disability) to 24 (severe disability), with a lower score indicating better function.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Units on a scale
  Screening (n=277) | 12.8 (5.22)
  Randomization Baseline (n=256) | 7.9 (5.14)
  Change from Screening (n=255) | -4.8 (4.95)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

43. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 2, 4, 8, and 12 (or Final Visit) in RMDQ Total Score
Description: as for outcome 42
Time Frame: Screening, Weeks 2, 4, 8, and 12
Population: ITT Population; imputation using the LOCF method for Week 12 only; Weeks 2, 4, 8 included observed cases. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a scale
  Week 2 (n=114,124) | -3.88 (0.423) | -4.93 (0.406)
  Week 4 (n=101,111) | -3.90 (0.467) | -4.60 (0.444)
  Week 8 (n=77,95) | -4.50 (0.514) | -3.92 (0.459)
  Week 12/ET (n=123,128) | -4.33 (0.440) | -4.26 (0.431)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Screening to Week 2; Test type: Superiority or Other; p = 0.0733, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = -1.05, 95% CI 2-sided [-2.20 to 0.10], Standard Error of Mean 0.584
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Screening to Week 4; Test type: Superiority or Other; p = 0.2783, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = -0.70, 95% CI 2-sided [-1.96 to 0.57], Standard Error of Mean 0.642
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Screening to Week 8; Test type: Superiority or Other; p = 0.3951, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = 0.58, 95% CI 2-sided [-0.77 to 1.93], Standard Error of Mean 0.684
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Screening to Week 12; Test type: Superiority or Other; p = 0.9063, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = 0.07, 95% CI 2-sided [-1.14 to 1.28], Standard Error of Mean 0.614

44. Secondary Outcome: Change From Randomization Baseline to the End of Double-Blind Weeks 2, 4, and 8 in RMDQ Total Score
Description: as for outcome 42
Time Frame: Randomization Baseline, Weeks 2, 4, and 8
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Units on a scale
  Week 2 (n=111,118) | 0.54 (0.334) | -0.19 (0.321)
  Week 4 (n=98,107) | 1.02 (0.420) | 0.32 (0.397)
  Week 8 (n=73,93) | -0.01 (0.471) | 0.41 (0.408)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted change from Baseline to Week 2; Test type: Superiority or Other; p = 0.1139, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Randomization Baseline score and final total daily dose of the Titration Period as covariates; Mean Difference (Net) = -0.74, 95% CI 2-sided [-1.65 to 0.18], Standard Error of Mean 0.463
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Baseline to Week 4; Test type: Superiority or Other; p = 0.2264, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -0.70, 95% CI 2-sided [-1.84 to 0.44], Standard Error of Mean 0.577
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Model-adjusted Change from Baseline to Week 8; Test type: Superiority or Other; p = 0.5074, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 0.41, 95% CI 2-sided [-0.81 to 1.63], Standard Error of Mean 0.619

45. Secondary Outcome: Percentage of Participants With Shift From Screening to Randomization Baseline in PGA of Low Back Pain by Category in Participants With Screening PGA Score of Very Good, Good, Fair, Poor, Very Poor
Description: Represents the score at Screening / score at Randomization Baseline in PGA of low back pain, a global evaluation that utilizes a 5-point Likert scale with a score of: 1 = very good, asymptomatic and no limitation of normal activities; 2 = good, mild symptoms, and no limitation of normal activities; 3 = fair, moderate symptoms and limitation to some normal activities; 4 = poor, severe symptoms and inability to carry out most normal activities; and a score of 5 = very poor; very severe symptoms, which were intolerable and inability to carry out all normal activities.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; percentage was based on the number of participants who had non-missing values at Randomization Baseline and Screening.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 277
Percentage of participants
  Very Good / Very Good | 0.4
  Very Good / Good | 2.9
  Very Good / Fair | 9.4
  Very Good / Poor | 2.9
  Very Good / Very Poor | 0.0
  Good / Very Good | 0.0
  Good / Good | 5.8
  Good / Fair | 29.2
  Good / Poor | 8.7
  Good / Very Poor | 1.4
  Fair / Very Good | 0.0
  Fair / Good | 2.5
  Fair / Fair | 22.0
  Fair / Poor | 10.5
  Fair / Very Poor | 1.4
  Poor / Very Good | 0.0
  Poor / Good | 0.4
  Poor / Fair | 2.2
  Poor / Poor | 0.4
  Poor / Very Poor | 0.0
  Very Poor / Very Good | 0.0
  Very Poor / Good | 0.0
  Very Poor / Fair | 0.0
  Very Poor / Poor | 0.0
  Very Poor / Very Poor | 0.0
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, Bowker's test of symmetry

46. Secondary Outcome: Percentage of Participants With Shift From Screening to the End of the Open-Label Titration Period in PGA of Low Back Pain by Category in Participants With Screening PGA Score of Very Good, Good, Fair, Poor, Very Poor
Description: Represents the score at Screening / score at to end of the titration period in PGA of low back pain, a global evaluation that utilizes a 5-point Likert scale with a score of: 1 = very good, asymptomatic and no limitation of normal activities; 2 = good, mild symptoms, and no limitation of normal activities; 3 = fair, moderate symptoms and limitation to some normal activities; 4 = poor, severe symptoms and inability to carry out most normal activities; and a score of 5 = very poor; very severe symptoms, which were intolerable and inability to carry out all normal activities.
Time Frame: Screening, Randomization Baseline, or Early Termination
Population: Titration Period Safety Population; percentage was based on the number of participants who had non-missing values at Randomization Baseline and Screening.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 368
Percentage of participants
  Very Good / Very Good | 0.3
  Very Good / Good | 2.7
  Very Good / Fair | 7.6
  Very Good / Poor | 2.2
  Very Good / Very Poor | 0.0
  Good / Very Good | 0.0
  Good / Good | 5.4
  Good / Fair | 25.0
  Good / Poor | 7.6
  Good / Very Poor | 1.1
  Fair / Very Good | 0.0
  Fair / Good | 2.7
  Fair / Fair | 27.2
  Fair / Poor | 10.6
  Fair / Very Poor | 1.4
  Poor / Very Good | 0.0
  Poor / Good | 0.3
  Poor / Fair | 3.0
  Poor / Poor | 2.2
  Poor / Very Poor | 0.3
  Very Poor / Very Good | 0.0
  Very Poor / Good | 0.0
  Very Poor / Fair | 0.0
  Very Poor / Poor | 0.3
  Very Poor / Very Poor | 0.3
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, Bowker's test of symmetry

47. Secondary Outcome: Percentage of Participants With Shift From Randomization Baseline to End of Double-Blind Week 4 in PGA of Low Back Pain by Category in Participants With Randomization Baseline PGA Score of Very Good, Good, Fair, Poor, Very Poor
Description: Represents the score at Randomization Baseline / score at Week 4 in PGA of low back pain, a global evaluation that utilizes a 5-point Likert scale with a score of: 1 = very good, asymptomatic and no limitation of normal activities; 2 = good, mild symptoms, and no limitation of normal activities; 3 = fair, moderate symptoms and limitation to some normal activities; 4 = poor, severe symptoms and inability to carry out most normal activities; and a score of 5 = very poor; very severe symptoms, which were intolerable and inability to carry out all normal activities.
Time Frame: Randomization Baseline, Week 4
Population: ITT Population; percentage was based on the number of participants who had non-missing values at Randomization Baseline and Week 4 for each treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 109 | 126
Percentage of participants
  Very Good / Very Good | 7.3 | 8.7
  Very Good / Good | 3.7 | 0.8
  Very Good / Fair | 0.9 | 0.0
  Very Good / Poor | 0.0 | 0.0
  Very Good / Very Poor | 0.0 | 0.0
  Good / Very Good | 5.5 | 6.3
  Good / Good | 24.8 | 27.8
  Good / Fair | 7.3 | 13.5
  Good / Poor | 0.0 | 0.0
  Good / Very Poor | 0.0 | 0.0
  Fair / Very Good | 0.9 | 1.6
  Fair / Good | 15.6 | 15.1
  Fair / Fair | 24.8 | 23.0
  Fair / Poor | 1.8 | 2.4
  Fair / Very Poor | 0.0 | 0.0
  Poor / Very Good | 0.9 | 0.0
  Poor / Good | 2.8 | 0.0
  Poor / Fair | 2.8 | 0.0
  Poor / Poor | 0.0 | 0.8
  Poor / Very Poor | 0.0 | 0.0
  Very Poor / Very Good | 0.0 | 0.0
  Very Poor / Good | 0.0 | 0.0
  Very Poor / Fair | 0.0 | 0.0
  Very Poor / Poor | 0.9 | 0.0
  Very Poor / Very Poor | 0.0 | 0.0
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.2211, Cochran-Mantel-Haenszel; Stratified by opioid stratum

48. Secondary Outcome: Percentage of Participants With Shift From Randomization Baseline to End of Double-Blind Week 8 in PGA of Low Back Pain by Category in Participants With Randomization Baseline PGA Score of Very Good , Good, Fair, Poor, Very Poor
Description: Represents the score at Randomization Baseline / score at Week 8 in PGA of low back pain, a global evaluation that utilizes a 5-point Likert scale with a score of: 1 = very good, asymptomatic and no limitation of normal activities; 2 = good, mild symptoms, and no limitation of normal activities; 3 = fair, moderate symptoms and limitation to some normal activities; 4 = poor, severe symptoms and inability to carry out most normal activities; and a score of 5 = very poor; very severe symptoms, which were intolerable and inability to carry out all normal activities.
Time Frame: Randomization Baseline, Week 8
Population: ITT Population; percentage was based on the number of participants who had non-missing values at Randomization Baseline and Week 8 for each treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 88 | 112
Percentage of participants
  Very Good / Very Good | 8.0 | 8.9
  Very Good / Good | 5.7 | 3.6
  Very Good / Fair | 0.0 | 1.8
  Very Good / Poor | 0.0 | 0.0
  Very Good / Very Poor | 0.0 | 0.0
  Good / Very Good | 5.7 | 8.0
  Good / Good | 25.0 | 23.2
  Good / Fair | 12.5 | 11.6
  Good / Poor | 0.0 | 0.9
  Good / Very Poor | 0.0 | 0.0
  Fair / Very Good | 3.4 | 0.9
  Fair / Good | 14.8 | 15.2
  Fair / Fair | 17.0 | 21.4
  Fair / Poor | 2.3 | 1.8
  Fair / Very Poor | 0.0 | 0.0
  Poor / Very Good | 0.0 | 0.0
  Poor / Good | 1.1 | 0.0
  Poor / Fair | 1.1 | 0.9
  Poor / Poor | 0.0 | 0.9
  Poor / Very Poor | 0.0 | 0.0
  Very Poor / Very Good | 0.0 | 0.0
  Very Poor / Good | 0.0 | 0.9
  Very Poor / Fair | 2.3 | 0.0
  Very Poor / Poor | 1.1 | 0.0
  Very Poor / Very Poor | 0.0 | 0.0
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.5767, Cochran-Mantel-Haenszel; Stratified by opioid stratum

49. Secondary Outcome: Satisfaction With Treatment at the End of Open-Label Titration Period for All Participants
Description: Satisfaction with treatment is a single-item self-rated instrument that measures the participant's overall satisfaction with the study drug during study participation on a 5-point likert scale ranging from 1 = Very dissatisfied to 5 = Very satisfied.
Time Frame: End of Open-Label Titration Period (Week 4, 5, or 6 or Early Termination)
Population: Titration Period Safety Population; percentage was based on the number of participants with non-missing response to treatment. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 369
Percentage of participants
  Very Dissatisfied (n=369) | 6.8
  Dissatisfied (n=369) | 7.0
  Neither Satisfied or Dissatisfied (n=369) | 11.7
  Satisfied (n=369) | 40.7
  Very Satisfied (n=369) | 33.9

50. Secondary Outcome: Satisfaction With Treatment at Randomization Baseline
Description: as for outcome 49
Time Frame: Randomization Baseline
Population: ITT Population; percentage was based on the number of participants with non-missing response to treatment. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 278
Percentage of participants
  Very Dissatisfied (n=278) | 5.4
  Dissatisfied (n=278) | 2.2
  Neither Satisfied or Dissatisfied (n=278) | 4.7
  Satisfied (n=278) | 46.0
  Very Satisfied (n=278) | 41.7

51. Secondary Outcome: Percentage of Participants Who Reported Being Satisfied/Very Satisfied With Treatment on the Satisfaction With Treatment Questionnaire During the Double-Blind Treatment Period
Description: Participants used an electronic tablet at the center to rate their overall treatment satisfaction with study drug during study participation using a 5-point categorical scale (1 = very dissatisfied, 2 = dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = satisfied, 5 = very satisfied).
Time Frame: Week 12 or Early Termination
Population: as for outcome 50
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 125 | 128
Percentage of participants
  Yes (n=125,128) | 59.2 | 79.7
  No (n=125,128) | 40.8 | 20.3
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by opioid stratum

52. Secondary Outcome: Change From Screening Period to the End of Open-Label Titration Period in Short Form-36v2 (SF-36v2) Health Survey Score
Description: SF-36v2 Health Survey is a self-administered questionnaire consisting of 36 questions, measuring 8 health aspects; physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception. These domains also combine to form two component summary scores evaluating mental health and physical health. The minimum score is 0 and the maximum score is 100. A higher scores indicates a better health state.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Score on a scale
  Physical Functioning (n=366) | 6.7 (8.96)
  Role-Physical (n=366) | 7.7 (9.48)
  Bodily Pain (n=366) | 9.8 (8.44)
  General Health (n=367) | 2.3 (6.54)
  Vitality (n=366) | 4.6 (8.98)
  Social Functioning (n=367) | 5.0 (11.01)
  Role-Emotional (n=367) | 3.4 (12.19)
  Mental Health (n=367) | 2.3 (8.76)
  Physical Component Score (n=364) | 8.2 (7.90)
  Mental Component Score (n=364) | 1.6 (10.05)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Physical Functioning; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Role-Physical; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Bodily Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for General Health; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 5: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Vitality; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 6: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Social Functioning; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 7: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Role-Emotional; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 8: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Mental Health; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 9: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Physical Component Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 10: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label Titration Period for Mental Component Score; Test type: Superiority or Other; p = 0.0026, t-test, 2 sided

53. Secondary Outcome: Change From Screening Period to Randomization Baseline in SF-36v2 Health Survey Score
Description: SF-36v2 Health Survey is a self-administered questionnaire consisting of 36 questions, measuring 8 health aspects; physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception. These domains also combine to form two component summary scores evaluating mental health and physical health. The minimum score is 0 and the maximum score is 100. A higher score indicate a better health state.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Score on a scale
  Physical Functioning (n=276) | 8.0 (8.90)
  Role-Physical (n=276) | 9.1 (9.40)
  Bodily Pain (n=276) | 11.6 (7.91)
  General Health (n=277) | 3.1 (6.65)
  Vitality (n=276) | 5.8 (9.08)
  Social Functioning (n=277) | 7.0 (10.27)
  Role-Emotional (n=277) | 4.7 (12.04)
  Mental Health (n=277) | 3.5 (8.29)
  Physical Component Score (n=274) | 9.6 (7.77)
  Mental Component Score (n=274) | 2.9 (9.69)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for Physical Functioning, Role-Physical, Bodily Pain, General Health, Vitality, Social Functioning, Role-Emotional, Mental Health, Physical Component Score, and Mental Component Score; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

54. Secondary Outcome: Change From Randomization Baseline to the End of Double-Blind Week 12 (or Final Visit) in SF-36v2 Health Survey
Description: as for outcome 53
Time Frame: Randomization Baseline, Week 12
Population: ITT Population; imputation using the LOCF method. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Score on a scale
  Physical Functioning (n=122,125) | -2.06 (0.681) | -1.44 (0.666)
  Role-Physical (n=124,126) | -2.56 (0.713) | -2.59 (0.701)
  Bodily Pain (n=124,127) | -5.07 (0.655) | -2.69 (0.643)
  General Health Perceptions (n=124,126) | -1.55 (0.545) | -2.10 (0.536)
  Vitality (n=123,127) | -1.62 (0.781) | -2.77 (0.762)
  Social Functioning (n=124,127) | -3.17 (0.748) | -1.69 (0.734)
  Role-Emotional (n=124,127) | -2.57 (0.963) | -3.44 (0.943)
  Mental Health (n=124,127) | -2.95 (0.711) | -2.93 (0.697)
  Physical Component Score (n=121,125) | -2.70 (0.635) | -1.68 (0.620)
  Mental Component Score (n=121,125) | -2.29 (0.767) | -2.98 (0.749)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Physical Functioning; Test type: Superiority or Other; p = 0.5181, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 0.62, 95% CI 2-sided [-1.26 to 2.49], Standard Error of Mean 0.952
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Role-Physical; Test type: Superiority or Other; p = 0.9733, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -0.03, 95% CI 2-sided [-2.00 to 1.93], Standard Error of Mean 0.998
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Bodily Pain; Test type: Superiority or Other; p = 0.0100, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 2.37, 95% CI 2-sided [0.57 to 4.18], Standard Error of Mean 0.914
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for General Health Perceptions; Test type: Superiority or Other; p = 0.4712, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -0.55, 95% CI 2-sided [-2.06 to 0.95], Standard Error of Mean 0.764
Statistical Analysis 5: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Vitality; Test type: Superiority or Other; p = 0.2898, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -1.16, 95% CI 2-sided [-3.30 to 0.99], Standard Error of Mean 1.091
Statistical Analysis 6: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Social Functioning; Test type: Superiority or Other; p = 0.1565, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 1.48, 95% CI 2-sided [-0.57 to 3.54], Standard Error of Mean 1.044
Statistical Analysis 7: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Role-Emotional; Test type: Superiority or Other; p = 0.5220, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -0.86, 95% CI 2-sided [-3.52 to 1.79], Standard Error of Mean 1.348
Statistical Analysis 8: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Mental Health; Test type: Superiority or Other; p = 0.9865, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 0.02, 95% CI 2-sided [-1.94 to 1.98], Standard Error of Mean 0.995
Statistical Analysis 9: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Physical Component Score; Test type: Superiority or Other; p = 0.2491, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 1.02, 95% CI 2-sided [-0.72 to 2.77], Standard Error of Mean 0.885
Statistical Analysis 10: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Randomization Baseline for Mental Component Score; Test type: Superiority or Other; p = 0.5219, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -0.69, 95% CI 2-sided [-2.80 to 1.43], Standard Error of Mean 1.073

55. Secondary Outcome: Change From Screening Period to End of Double-Blind Week 12 (or Final Visit) in SF-36v2 Health Survey
Description: as for outcome 53
Time Frame: Screening, Week 12
Population: as for outcome 54
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Score on a scale
  Physical Functioning (n=123,126) | 5.32 (0.794) | 6.84 (0.787)
  Role-Physical (n=125,127) | 5.68 (0.805) | 6.78 (0.802)
  Bodily Pain (n=125,127) | 6.39 (0.747) | 8.78 (0.743)
  General Health Perceptions (n=125,126) | 1.28 (0.611) | 1.07 (0.609)
  Vitality (n=125,127) | 3.46 (0.798) | 3.01 (0.794)
  Social Functioning (n=125,127) | 3.58 (0.771) | 5.57 (0.768)
  Role-Emotional (n=125,127) | 0.99 (0.979) | 1.22 (0.975)
  Mental Health (n=125,127) | 0.09 (0.752) | 0.47 (0.748)
  Physical Component Score (n=123,126) | 6.42 (0.721) | 8.09 (0.715)
  Mental Component Score (n=123,126) | -0.44 (0.816) | -0.45 (0.808)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Physical Functioning; Test type: Superiority or Other; p = 0.1731, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 1.52, 95% CI 2-sided [-0.67 to 3.71], Standard Error of Mean 1.111
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Role-Physical; Test type: Superiority or Other; p = 0.3290, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 1.10, 95% CI 2-sided [-1.12 to 3.32], Standard Error of Mean 1.127
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Bodily Pain; Test type: Superiority or Other; p = 0.0232, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 2.39, 95% CI 2-sided [0.33 to 4.45], Standard Error of Mean 1.047
Statistical Analysis 4: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for General Health Perceptions; Test type: Superiority or Other; p = 0.8139, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -0.20, 95% CI 2-sided [-1.89 to 1.49], Standard Error of Mean 0.858
Statistical Analysis 5: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Vitality; Test type: Superiority or Other; p = 0.6878, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -0.45, 95% CI 2-sided [-2.65 to 1.75], Standard Error of Mean 1.117
Statistical Analysis 6: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Social Functioning; Test type: Superiority or Other; p = 0.0658, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 2.00, 95% CI 2-sided [-0.13 to 4.12], Standard Error of Mean 1.080
Statistical Analysis 7: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Role-Emotional; Test type: Superiority or Other; p = 0.8670, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 0.23, 95% CI 2-sided [-2.48 to 2.94], Standard Error of Mean 1.374
Statistical Analysis 8: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Mental Health; Test type: Superiority or Other; p = 0.7259, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 0.37, 95% CI 2-sided [-1.71 to 2.45], Standard Error of Mean 1.056
Statistical Analysis 9: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Physical Component Score; Test type: Superiority or Other; p = 0.0989, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = 1.67, 95% CI 2-sided [-0.32 to 3.65], Standard Error of Mean 1.007
Statistical Analysis 10: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Difference between treatment groups in change from Screening for Mental Component Score; Test type: Superiority or Other; p = 0.9969, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -0.00, 95% CI 2-sided [-2.25 to 2.25], Standard Error of Mean 1.142

56. Secondary Outcome: Change From Screening Period to the End of Open-Label Titration Period in Participant Assessment of Overall Health State Using the EuroQol 5-Dimensions (EQ-5D) Summary Index
Description: The EQ 5D Health Questionnaire is a self completion standardized instrument for use as a measure of health-related quality of life in terms of a single index value or utility score that consisted of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which was rated on a 3-point response scale (no problems/some or moderate problems/extreme problems), and the scores are combined to form a single index utility value between 0 and 1 with higher scores indicating better health.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Score on a scale
  Screening (n=400) | 0.68 (0.174)
  End of Open-Label (n=354) | 0.80 (0.134)
  Change from Screening (n=346) | 0.12 (0.174)
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

57. Secondary Outcome: Change From Screening Period to the End of Open-Label Titration Period in Participant Assessment of Overall Health State Using the EQ-5D VAS
Description: The EQ-5D consists of a standard vertical 20cm visual analogue scale (EQ VAS), for recording a participant's rating for their current health related quality of life state; the scale went from 0 (worst imaginable health state) to 100 (best imaginable health state). Participants were asked to draw a line on the scale to indicate how good or bad your own health is today, in your opinion.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Score on a scale
  Screening (n=406) | 66.23 (18.277)
  End of Open-Label (n=367) | 74.69 (18.204)
  Change from Screening (n=364) | 8.16 (19.398)
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

58. Secondary Outcome: Change From Screening Period to Randomization Baseline in Participant Assessment of Overall Health State Using the EQ-5D Summary Index
Description: Self-completion standardized instrument for use as a measure of health-related quality of life in terms of a single index value or utility score that consisted of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which was rated on a 3-point response scale (no problems/some or moderate problems/extreme problems), and the scores are combined to form a single index utility value between 0 and 1 with higher scores indicating better health
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Score on a scale
  Screening (n=272) | 0.68 (0.178)
  Randomization Baseline (n=267) | 0.82 (0.120)
  Change from Screening (n=260) | 0.14 (0.177)
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

59. Secondary Outcome: Change From Screening Period to Randomization Baseline in Participant Assessment of Overall Health State Using the EQ-5D VAS
Description: as for outcome 57
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Score on a scale
  Screening (n=279) | 67.02 (18.518)
  Randomization Baseline (n=276) | 76.85 (17.407)
  Change from Screening (n=275) | 9.84 (19.692)
Statistical Analysis 1: Comparison: Open ALO-02; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

60. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Week 12 (or Final Visit) in Participant Assessment of Overall Health State Using EQ-5D Summary Index
Description: as for outcome 58
Time Frame: Randomization Baseline, Week 12
Population: as for outcome 54
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 118 | 115
Score on a scale | -0.061 (0.0118) | -0.029 (0.0120)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.0605, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Randomization Baseline score and final total daily dose of study drug during the Titration Period as covariates; Mean Difference (Net) = 0.032, 95% CI 2-sided [-0.001 to 0.065], Standard Error of Mean 0.0168

61. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Week 12 (or Final Visit) in Participant Assessment of Overall Health State Using the EQ-5D VAS
Description: as for outcome 57
Time Frame: Randomization Baseline, Week 12
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 122 | 126
Score on a scale | -3.61 (1.432) | -2.89 (1.401)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.7196, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors; Randomization Baseline score and final total daily dose of study drug during the Titration Period as covariates; Mean Difference (Net) = 0.72, 95% CI 2-sided [-3.22 to 4.66], Standard Error of Mean 1.999

62. Secondary Outcome: Change From Screening Period to End of Double-Blind Week 12 (or Final Visit) in Participant Assessment of Overall Health State Using EQ-5D Summary Index
Description: as for outcome 58
Time Frame: Screening, Week 12
Population: as for outcome 54
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 121 | 117
Score on a scale | 0.085 (0.0121) | 0.106 (0.0124)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.2280, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = 0.021, 95% CI 2-sided [-0.013 to 0.055], Standard Error of Mean 0.0172

63. Secondary Outcome: Change From Screening Period to End of Double-Blind Week 12 (or Final Visit) in Participant Assessment of Overall Health State Using EQ-5D VAS
Description: as for outcome 57
Time Frame: Screening, Week 12
Population: as for outcome 54
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 124 | 127
Score on a scale | 4.75 (1.465) | 7.01 (1.454)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Test type: Superiority or Other; p = 0.2701, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariate; Mean Difference (Net) = 2.26, 95% CI 2-sided [-1.77 to 6.30], Standard Error of Mean 2.048

64. Secondary Outcome: Change From Screening Period to End of Open-Label in Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP): % Work Time Missed, % Impairment, % Overall Work Impairment, % Activity Impairment Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment /absenteeism+presenteeism); and activity impairment.
  * work time missed - a measure of absenteeism, calculated as work time missed due to health problem (question 2) as a proportion of hours actually worked (question 4).
  * impairment while working - a measure of presenteeism, the degree to which health problem impacted work (question 5).
  * overall work impairment - a measure of overall work productivity loss due to health problem (absenteeism+presenteeism).
  * activity impairment - a measure of the degree to which health problem has affected ability to do regular activities other than work at a job (question 6). Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Percentage
  Percent Work Time Missed (n=119) | -1.3 (16.66)
  Percent Impairment While Working (n=112) | -22.4 (26.95)
  Percent Overall Work Impairment (n=110) | -21.6 (29.83)
  Percent Activity Impairment (n=363) | -27.2 (24.45)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label for % Work Time Missed due to Low Back Pain; Test type: Superiority or Other; p = 0.3822, t-test, 2 sided
Statistical Analysis 2: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label for % Impairment while Working due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label for % Overall Work Impairment due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Open ALO-02; Change from Screening Period value to End of Open-Label for % Activity Impairment due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

65. Secondary Outcome: Change From Screening Period to Randomization Baseline in WPAI:SHP: Percent Work Time Missed, Percent Impairment, Percent Overall Work Impairment, Percent Activity Impairment Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism+presenteeism); and activity impairment.
  * work time missed - a measure of absenteeism, calculated as work time missed due to health problem (question 2) as a proportion of hours actually worked (question 4).
  * impairment while working - a measure of presenteeism, the degree to which health problem impacted work (question 5).
  * overall work impairment - a measure of overall work productivity loss due to health problem (absenteeism+presenteeism).
  * activity impairment - a measure of the degree to which health problem has affected ability to do regular activities other than work at a job (question 6).
  Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Percentage
  Percent Work Time Missed (n=91) | -4.9 (14.37)
  Percent Impairment While Working (n=86) | -25.9 (27.24)
  Percent Overall Work Impairment (n=85) | -26.9 (27.76)
  Percent Activity Impairment (n=273) | -32.0 (23.96)
Statistical Analysis 1: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for % Work Time Missed due to Low Back Pain; Test type: Superiority or Other; p = 0.0017, t-test, 2 sided
Statistical Analysis 2: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for % Impairment while Working due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 3: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for % Overall Work Impairment due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Open ALO-02; Change from Screening Period value to Randomization Baseline for % Activity Impairment due to Low Back Pain; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

66. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Work Time Missed Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism+presenteeism); and activity impairment.
  % work time missed - a measure of absenteeism, calculated as work time missed due to health problem (question 2) as a proportion of hours actually worked (question 4).
  Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: ITT Population; imputation by the LOCF method was used for Week 12 (or Final Visit) only; Weeks 4 and 8 were based on observed cases. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 44 | 56
Percentage
  Week 4 (n=36,44) | 3.54 (2.213) | -0.77 (1.906)
  Week 8 (n=25,41) | 4.29 (3.507) | 1.41 (2.592)
  Week 12/ET (n=40,50) | 6.49 (3.108) | 3.72 (2.675)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.1389, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -4.31, 95% CI 2-sided [-10.06 to 1.43], Standard Error of Mean 2.883
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.5094, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -2.88, 95% CI 2-sided [-11.56 to 5.80], Standard Error of Mean 4.340
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.4944, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -2.77, 95% CI 2-sided [-10.81 to 5.26], Standard Error of Mean 4.043

67. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Impairment Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism+presenteeism); and activity impairment.
  % impairment while working - a measure of presenteeism, the degree to which health problem impacted work (question 5).
  Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 42 | 54
Percentage
  Week 4 (n=30,42) | 5.22 (3.366) | -1.54 (2.734)
  Week 8 (n=21,37) | 3.63 (4.318) | -1.36 (3.027)
  Week 12/ET (n=35,46) | 6.77 (3.475) | 4.39 (2.918)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.1201, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -6.76, 95% CI 2-sided [-15.33 to 1.81], Standard Error of Mean 4.295
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.3497, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -4.99, 95% CI 2-sided [-15.60 to 5.62], Standard Error of Mean 5.288
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.6008, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -2.38, 95% CI 2-sided [-11.41 to 6.65], Standard Error of Mean 4.532

68. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Overall Work Impairment Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism+presenteeism); and activity impairment.
  % overall work impairment - a measure of overall work productivity loss due to health problem (absenteeism+presenteeism).
  Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 42 | 53
Percentage
  Week 4 (n=30,42) | 5.31 (3.894) | -2.03 (3.147)
  Week 8 (n=21,37) | 8.69 (5.276) | -0.66 (3.666)
  Week 12/ET (n=35,46) | 10.85 (4.266) | 5.71 (3.575)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.1458, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -7.34, 95% CI 2-sided [-17.29 to 2.62], Standard Error of Mean 4.986
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.1558, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -9.35, 95% CI 2-sided [-22.38 to 3.68], Standard Error of Mean 6.496
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.3604, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -5.14, 95% CI 2-sided [-16.25 to 5.98], Standard Error of Mean 5.582

69. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Activity Impairment Due to Low Back Pain
Description: A self-reported measure of work productivity and impairment that yields 4 scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on the job effectiveness); work productivity loss (overall work impairment/absenteeism+presenteeism); and activity impairment.
  % activity impairment - a measure of the degree to which health problem has affected ability to do regular activities other than work at a job (question 6). Each score is expressed as a percentage (0-100%) with higher numbers indicating greater impairment and less productivity.
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 131 | 144
Percentage
  Week 4 (n=108,125) | 6.23 (1.768) | 1.98 (1.626)
  Week 8 (n=85,112) | 2.05 (2.044) | 3.05 (1.752)
  Week 12/ET (n=128,135) | 10.56 (1.818) | 6.41 (1.758)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.0768, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -4.25, 95% CI 2-sided [-8.95 to 0.46], Standard Error of Mean 2.389
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.7109, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = 1.00, 95% CI 2-sided [-4.30 to 6.29], Standard Error of Mean 2.684
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.1031, ANCOVA — [p-value comment as in outcome 44, analysis 1]; Mean Difference (Net) = -4.15, 95% CI 2-sided [-9.14 to 0.85], Standard Error of Mean 2.536

70. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Work Time Missed Due to Low Back Pain
Description: as for outcome 66
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 46 | 58
Percentage
  Week 4 (n=36,43) | -0.09 (2.147) | -4.82 (1.911)
  Week 8 (n=24,40) | -1.42 (2.785) | -3.01 (2.123)
  Week 12/ET (n=40,49) | -1.00 (2.612) | -2.09 (2.307)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.0926, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -4.73, 95% CI 2-sided [-10.26 to 0.80], Standard Error of Mean 2.776
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.6437, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -1.59, 95% CI 2-sided [-8.42 to 5.24], Standard Error of Mean 3.414
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.7480, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -1.09, 95% CI 2-sided [-7.84 to 5.65], Standard Error of Mean 3.391

71. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Impairment Due to Low Back Pain
Description: as for outcome 67
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 47 | 56
Percentage
  Week 4 (n=33,42) | -18.65 (3.614) | -31.03 (3.151)
  Week 8 (n=22,37) | -16.43 (4.374) | -29.37 (3.263)
  Week 12/ET (n=38,46) | -16.18 (3.642) | -25.38 (3.242)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.0098, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -12.38, 95% CI 2-sided [-21.68 to -3.07], Standard Error of Mean 4.666
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.0186, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -12.94, 95% CI 2-sided [-23.63 to -2.25], Standard Error of Mean 5.336
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.0581, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -9.20, 95% CI 2-sided [-18.72 to 0.32], Standard Error of Mean 4.785

72. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Overall Work Impairment Due to Low Back Pain
Description: as for outcome 68
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 46 | 56
Percentage
  Week 4 (n=32,41) | -19.84 (3.992) | -32.40 (3.470)
  Week 8 (n=21,37) | -15.21 (4.933) | -29.37 (3.608)
  Week 12/ET (n=37,46) | -15.16 (4.268) | -25.51 (3.759)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.0177, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -12.56, 95% CI 2-sided [-22.87 to -2.25], Standard Error of Mean 5.168
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.0219, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -14.16, 95% CI 2-sided [-26.19 to -2.14], Standard Error of Mean 5.998
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.0679, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -10.35, 95% CI 2-sided [-21.47 to 0.78], Standard Error of Mean 5.589

73. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in WPAI:SHP Percent Activity Impairment Due to Low Back Pain
Description: as for outcome 69
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 66
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 133 | 145
Percentage
  Week 4 (n=109,125) | -23.75 (1.960) | -31.24 (1.829)
  Week 8 (n=87,112) | -25.25 (2.279) | -29.87 (2.005)
  Week 12/ET (n=130,136) | -18.62 (2.025) | -26.81 (1.981)
Statistical Analysis 1: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 4; Test type: Superiority or Other; p = 0.0052, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -7.50, 95% CI 2-sided [-12.72 to -2.27], Standard Error of Mean 2.654
Statistical Analysis 2: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 8; Test type: Superiority or Other; p = 0.1249, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -4.62, 95% CI 2-sided [-10.54 to 1.29], Standard Error of Mean 2.999
Statistical Analysis 3: Comparison: ALO-02 To Placebo vs ALO-02 To ALO-02; Week 12/ET; Test type: Superiority or Other; p = 0.0040, ANCOVA — Treatment and prior pain analgesic (opioid or non-opioid) as categorical factors and the Screening score as covariates; Mean Difference (Net) = -8.19, 95% CI 2-sided [-13.74 to -2.64], Standard Error of Mean 2.818

74. Secondary Outcome: Percentage of Participants With Shift From Screening Period to End of Open-Label Titration Period in Hospitalization Because of Low Back Pain as Assessed Using the Healthcare Resource Use (HRU) Questionnaire
Description: Question 3a = In the past 4 weeks, have you been hospitalized due to chronic low back pain or any medication used for chronic low back pain?
Time Frame: Screening, Week 6 (or Early Termination)
Population: Titration Period Safety Population; the denominator for the percentage calculation is the number of participants who had both Screening value and End of Open-Label value.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 362
Percentage of participants
  Yes/Yes | 0.3
  Yes/No | 0.8
  No/Yes | 2.5
  No/No | 96.4

75. Secondary Outcome: Percentage of Participants With Shift From Screening Period to Randomization Baseline in Hospitalization Because of Low Back Pain as Assessed Using the HRU Questionnaire
Description: as for outcome 74
Time Frame: Screening, Randomization Baseline
Population: ITT Population; the denominator for the percentage calculation is the number of participants who had both Screening value and Randomization Baseline value.
Measure: Number; unit: Percentage of participants
Arm/Group | Open ALO-02
Number analyzed (Participants) | 272
Percentage of participants
  Yes/Yes | 0.4
  Yes/No | 1.1
  No/Yes | 2.9
  No/No | 95.6

76. Secondary Outcome: Change From Screening to Randomization Baseline in HRU Questionnaire: Number of Office Visits Directly Related or Any Medication Used for Chronic Low Back Pain
Description: Question 1: number of office visits directly related to chronic low back pain or any medication used for chronic low back pain.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Number of visits
  Screening (n=257) | 11.4 (38.97)
  Randomization Baseline (n=247) | 5.6 (21.84)
  Change from Screening (n=234) | -4.7 (39.19)

77. Secondary Outcome: Change From Screening to Randomization Baseline in HRU Questionnaire: Money Spent on Physical Treatments in Past 4 Weeks
Description: Question 2: Money (dollars) spent out-of-pocket on physical treatments in the past 4 weeks to manage chronic low back pain
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Dollars
  Screening (n=264) | 84.7 (418.06)
  Randomization Baseline (n=260) | 51.8 (360.94)
  Change from Screening (n=248) | -41.8 (522.53)

78. Secondary Outcome: Change From Screening to Randomization Baseline in HRU Questionnaire: Nights Stayed in Hospital
Description: Question 3b: nights stayed in the hospital, if answer to Q3a was yes.
Time Frame: Screening, Randomization Baseline
Population: ITT Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 280
Number of days
  Screening (n=9) | 0.1 (0.33)
  Randomization Baseline (n=3) | 0.0 (0.00)
  Change from Screening (n=1) | 0.0 (NA) — Standard Deviation not applicable as n=1

79. Secondary Outcome: Change From Screening to End of Open-Label Titration Period in HRU Questionnaire: Number of Office Visits Directly Related or Any Medication Used for Chronic Low Back Pain
Description: as for outcome 76
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Number of visits
  Screening (n=373) | 8.8 (33.07)
  Randomization Baseline (n=325) | 5.4 (20.58)
  Change from Screening (n=308) | -3.0 (35.29)

80. Secondary Outcome: Change From Screening to End of Open-Label Titration Period in HRU Questionnaire: Money Spent on Physical Treatments in Past 4 Weeks
Description: as for outcome 77
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Dollars
  Screening (n=388) | 104.1 (605.48)
  Randomization Baseline (n=343) | 88.0 (674.20)
  Change from Screening (n=329) | -28.3 (548.03)

81. Secondary Outcome: Change From Screening to End of Open-Label Titration Period in HRU Questionnaire: Nights Stayed in Hospital
Description: Question 3b: nights stayed in the hospital, if answer to Q3a was yes.
Time Frame: Screening, Week 6 (or Early Termination)
Population: as for outcome 35
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
Number of days
  Screening (n=9) | 0.1 (0.33)
  Randomization Baseline (n=3) | 0.0 (0.00)
  Change from Screening (n=1) | 0.0 (NA) — Standard Deviation not applicable as n=1

82. Secondary Outcome: Percentage of Participants With Shift From Randomization Baseline to End of Double-Blind Weeks 4, 8, and 12 (or Final Visit) in Hospitalization Because of Low Back Pain as Assessed Using the HRU Questionnaire
Description: as for outcome 74
Time Frame: Randomization Baseline, Weeks 4, 8, and 12 (or Early Termination)
Population: ITT Population; the denominator for the percentage calculation is the number of participants who had both Randomization Baseline value and Post Randomization value for each treatment and visit. Imputation using the LOCF method.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Percentage of participants
  Yes/Yes Week 4 (n=108, 123) | 0.0 | 0.0
  Yes/No Week 4 (n=108, 123) | 3.7 | 0.8
  No/Yes Week 4 (n=108, 123) | 1.9 | 0.0
  No/No Week 4 (n=108, 123) | 94.4 | 99.2
  Yes/Yes Week 8 (n=85, 110) | 0.0 | 0.0
  Yes/No Week 8 (n=85, 110) | 1.2 | 0.9
  No/Yes Week 8 (n=85, 110) | 2.4 | 0.0
  No/No Week 8 (n=85, 110) | 96.5 | 99.1
  Yes/Yes Week12/ET (n=129, 134) | 0.0 | 0.0
  Yes/No Week12/ET (n=129, 134) | 3.1 | 0.0
  No/Yes Week12/ET (n=129, 134) | 1.6 | 0.7
  No/No Week 12/ET (n=129, 134) | 95.3 | 99.3

83. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Number of Office Visits Related to or Medications Used for Chronic Low Back Pain
Description: as for outcome 76
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Number of visits
  Randomization Baseline (n=118,129) | 4.4 (18.10) | 6.6 (24.80)
  Week 4 (n=100,110) | 6.5 (24.35) | 5.3 (37.99)
  Change from Baseline at Week 4 (n=95,106) | 0.1 (24.17) | -3.1 (46.85)
  Week 8 (n=79,103) | 22.8 (179.55) | 3.3 (13.46)
  Change from Baseline at Week 8 (n=74,100) | -1.2 (20.35) | -2.6 (24.31)
  Week 12/ET (n=121,128) | 19.2 (153.80) | 4.2 (15.38)
  Change from Baseline at Week 12/ET (n=112,119) | -0.3 (24.90) | -4.1 (27.74)

84. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Money Spent on Treatments
Description: as for outcome 77
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: ITT Population, imputation using the LOCF method. n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Dollars
  Randomization Baseline (n=124,136) | 96.4 (518.89) | 11.3 (33.77)
  Week 4 (n=104,119) | 19.9 (90.26) | 15.0 (78.59)
  Change from Baseline at Week 4 (n=99,117) | -24.7 (222.07) | 4.4 (79.92)
  Week 8 (n=81,106) | 146.2 (1113.58) | 16.7 (54.33)
  Change from Baseline at Week 8 (n=76,105) | -0.1 (71.11) | 7.5 (42.52)
  Week 12/ET (n=125,133) | 113.0 (913.41) | 29.3 (177.85)
  Change from Baseline at Week 12/ET (n=119,128) | -47.8 (461.95) | 20.0 (180.70)

85. Secondary Outcome: Change From Randomization Baseline to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Nights Spent in Hospital
Description: Question 3b: nights stayed in the hospital
Time Frame: Randomization Baseline, Weeks 4, 8, and 12
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: Number of nights
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Number of nights
  Randomization Baseline (n=1,2) | 0.0 (NA) — Standard deviation not applicable as n=1 | 0.0 (0.00)
  Week 4 (n=4,0) | 0.3 (0.5) | NA (NA) — Mean and standard deviation not applicable as n=0
  Change from Baseline at Week 4 (n=0,0) | NA (NA) — Mean and standard deviation not applicable as n=0 | NA (NA) — Mean and standard deviation not applicable as n=0
  Week 8 (n=1,1) | 99.0 (NA) — Standard deviation not applicable as n=1 | 0.0 (NA) — Standard deviation not applicable as n=1
  Change from Baseline at Week 8 (n=0,0) | NA (NA) — Mean and standard deviation not applicable as n=0 | NA (NA) — Mean and standard deviation not applicable as n=0
  Week 12/ET (n=4,1) | 24.8 (49.50) | 0.0 (NA) — standard deviation not applicable as n=1
  Change from Baseline at Week 12/ET (n=0,0) | NA (NA) — Mean and standard deviation not applicable as n=0 | NA (NA) — Mean and standard deviation not applicable as n=0

86. Secondary Outcome: Percentage of Participants With Shift From Screening Period to the End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in Hospitalization Because of Low Back Pain as Assessed Using the HRU Questionnaire
Description: as for outcome 74
Time Frame: Screening, Weeks 4, 8, and 12
Population: ITT Population; the denominator for the percentage calculation is the number of participants who had both Screening value and Post Screening value for each treatment and visit. Imputation using the LOCF method.
Measure: Number; unit: Percentage of participants
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Percentage of participants
  Yes/Yes Week 4 (n=109,124) | 0.9 | 0.0
  Yes/No Week 4 (n=109,124) | 2.8 | 0.8
  No/Yes Week 4 (n=109,124) | 2.8 | 1.6
  No/No Week 4 (n=109,124) | 93.6 | 97.6
  Yes/Yes Week 8 (n=86,111) | 0.0 | 0.0
  Yes/No Week 8 (n=86, 111) | 1.2 | 0.9
  No/Yes Week 8 (n=86, 111) | 2.3 | 1.8
  No/No Week 8 (n=86, 111) | 96.5 | 97.3
  Yes/Yes Week 12/ET (n=130,136) | 0.8 | 0.0
  Yes/No Week 12/ET (n=130,136) | 2.3 | 0.0
  No/Yes Week 12/ET (n=130,136) | 3.8 | 2.2
  No/No Week 12/ET (n=130,136) | 93.1 | 97.8

87. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Number of Office Visits Related or Medication Used for Chronic Low Back Pain
Description: as for outcome 76
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: Number of visits
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Number of visits
  Screening (n=121,136) | 8.8 (33.76) | 13.7 (43.07)
  Week 4 (n=100,110) | 6.5 (24.35) | 5.3 (37.99)
  Change from Screening at Week 4 (n=94,106) | 0.8 (28.99) | -7.6 (58.56)
  Week 8 (n=79,103) | 22.8 (179.55) | 3.3 (13.46)
  Change from Screening at Week 8 (n=73,100) | 16.7 (188.74) | -10.4 (44.61)
  Week 12/ET (n=121,128) | 19.2 (153.80) | 4.2 (15.38)
  Change from Screening at Week 12/ET (n=114,123) | 13.2 (159.55) | -7.3 (41.80)

88. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Money Spent on Treatment for Chronic Low Back Pain
Description: as for outcome 77
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Dollars
  Screening (n=126,138) | 83.6 (277.98) | 85.6 (514.80)
  Week 4 (n=104,119) | 19.9 (90.26) | 15.0 (78.59)
  Change from Screening at Week 4 (n=100,114) | -79.8 (315.79) | -80.3 (497.56)
  Week 8 (n=81,106) | 146.2 (1113.58) | 16.7 (54.33)
  Change from Screening at Week 8 (n=78,103) | 56.9 (1174.87) | -84.5 (593.49)
  Week 12/ET (n=125,133) | 113.0 (913.41) | 29.3 (177.85)
  Change from Screening at Week 12/ET (n=120,128) | 32.1 (944.71) | -58.1 (563.65)

89. Secondary Outcome: Change From Screening Period to End of Double-Blind Weeks 4, 8 and 12 (or Final Visit) in HRU Questionnaire: Nights in Hospital for Chronic Low Back Pain
Description: Question 3b: nights stayed in the hospital
Time Frame: Screening, Weeks 4, 8, and 12
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: Number of nights
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
Number of nights
  Screening (n=6,3) | 0.0 (0.00) | 0.3 (0.58)
  Week 4 (n=4,0) | 0.3 (0.50) | NA (NA) — Mean and Standard deviation not applicable as n=0
  Change from Screening at Week 4 (n=1,0) | 0.0 (NA) — Standard deviation not applicable as n=1 | NA (NA) — Mean and Standard deviation not applicable as n=0
  Week 8 (n=1,1) | 99.0 (NA) — Standard deviation not applicable as n=1 | 0.0 (NA) — Standard deviation not applicable as n=1
  Change from Screening at Week 8 (n=0,0) | NA (NA) — Mean and Standard deviation not applicable as n=0 | NA (NA) — Mean and Standard deviation not applicable as n=0
  Week 12/ET (n=4,1) | 24.8 (49.50) | 0.0 (NA) — Standard deviation not applicable as n=1
  Change from Screening at Week 12/ET (n=1,0) | 0.0 (NA) — Standard deviation not applicable as n=1 | NA (NA) — Mean and Standard deviation not applicable as n=0

90. Secondary Outcome: Mean Oxycodone Average Daily Dose During the Open-Label Titration Period
Time Frame: Open-Label Period
Population: Titration Period Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
mg | 45.8 (22.61)

91. Secondary Outcome: Mean Oxycodone Duration of Titration During the Open-Label Titration Period
Time Frame: Open-Label Period
Population: Titration Period Safety Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
days | 31.0 (12.24)

92. Secondary Outcome: Median Oxycodone Average Daily Dose During the Open-Label Titration Period
Time Frame: Open-Label Period
Population: Titration Period Safety Population
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
mg | 42.3 (22.61) [16 to 163]

93. Secondary Outcome: Median Oxycodone Duration of Titration During the Open-Label Titration Period
Time Frame: Open-Label Period
Population: Titration Period Safety Population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
days | 35.0 (12.24) [1 to 56]

94. Secondary Outcome: Mean Oxycodone Average Daily Dose During the Double-Blind Treatment Period
Time Frame: Double-Blind Period
Population: Double-Blind Safety Population
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
mg | 70.1 (33.67) | 63.6 (34.02)

95. Secondary Outcome: Mean Oxycodone Duration of Treatment During the Double-Blind Treatment Period
Time Frame: Double-Blind Period
Population: Double-Blind Safety Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
days | 62.7 (30.20) | 70.9 (27.80)

96. Secondary Outcome: Median Oxycodone Average Daily Dose During the Double-Blind Treatment Period
Time Frame: Double-Blind Period
Population: Double-Blind Safety Population
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
mg | 60.0 [20 to 152] | 59.6 [19 to 160]

97. Secondary Outcome: Median Oxycodone Duration of Treatment During the Double-Blind Treatment Period
Time Frame: Double-Blind Period
Population: Double-Blind Safety Population
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
days | 84.0 [5 to 94] | 85.0 [1 to 102]

98. Secondary Outcome: Oxycodone and Noroxycodone Observed Steady-State Plasma Concentration During the Titration Period
Description: Observed steady-state plasma concentration (Cobs) of oxycodone and noroxycodone.
Time Frame: Blood samples were taken within +/-4 hours of the morning dose of ALO-02 at Week 6/Early Termination, Randomization Baseline
Population: Titration Period Safety Population; participants assessed at Week 6 had not been randomized to the Double-Blind Period; participants assessed at Randomization Baseline had been randomized to the Double-Blind Period.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
ng/mL
  Oxycodone at Week 6/ET (n=77) | 14.1 (22.27)
  Oxycodone at Randomization Baseline (n=267) | 26.4 (28.84)
  Noroxycodone at Week 6/ET (n=77) | 15.5 (26.50)
  Noroxycodone at Randomization Baseline (n=267) | 29.9 (42.04)

99. Secondary Outcome: Naltrexone and 6-β-naltrexol Observed Steady-State Plasma Concentration During the Titration Period
Description: Cobs of naltrexone and 6-β-naltrexol
Time Frame: as for outcome 98
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Open ALO-02
Number analyzed (Participants) | 410
pg/mL
  Naltrexone at Week 6/ET (n=77) | 4.6 (19.02)
  Naltrexone at Randomization Baseline (n=266) | 14.6 (81.73)
  6-β-naltrexol at Week 6/ET (n=77) | 82.0 (305.91)
  6-β-naltrexol at Randomization Baseline (n=266) | 154.1 (595.80)

100. Secondary Outcome: Oxycodone and Noroxycodone Observed Steady-State Plasma Concentration During the Double-Blind Treatment Period
Description: Observed steady-state plasma concentration (Cobs) of oxycodone and noroxycodone
Time Frame: Blood samples were taken within +/-4 hours of the morning dose of study drug at Randomization Baseline, Weeks 4, 8, and 12
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
ng/mL
  Oxycodone at Baseline (n=127,140) | 27.0 (29.06) | 25.9 (28.73)
  Oxycodone at Week 4 (n=0,116) | NA (NA) — Mean and standard deviation not applicable as n=0 | 23.3 (26.90)
  Oxycodone at Week 8 (n=0,107) | NA (NA) — Mean and standard deviation not applicable as n=0 | 23.1 (23.83)
  Oxycodone at Week 12/ET (n=1,137) | 0.0 (NA) — Standard deviation not applicable as n=1 | 22.6 (26.98)
  Noroxycodone at Baseline (n=127,140) | 33.1 (48.84) | 27.1 (34.67)
  Noroxycodone at Week 4 (n=0,116) | NA (NA) — Mean and standard deviation not applicable as n=0 | 25.5 (40.54)
  Noroxycodone at Week 8 (n=0,107) | NA (NA) — Mean and standard deviation not applicable as n=0 | 26.2 (34.38)
  Noroxycodone at Week 12/ET (n=1,137) | 0.0 (NA) — Standard deviation not applicable as n=0 | 26.3 (40.67)

101. Secondary Outcome: Naltrexone and 6-β-naltrexol Observed Steady-State Plasma Concentration During the Double Blind Treatment Period
Description: Observed steady-state plasma concentration (Cobs) of naltrexone and 6-β-naltrexol
Time Frame: as for outcome 100
Population: Double-Blind Safety Population; n=number of participants analyzed for the given parameter at the specified timepoint.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | ALO-02 To Placebo | ALO-02 To ALO-02
Number analyzed (Participants) | 134 | 146
pg/mL
  Naltrexone at Baseline (n=127,139) | 24.9 (116.41) | 5.3 (16.48)
  Naltrexone at Week 4 (n=3,115) | 0.0 (0.0) | 3.4 (14.65)
  Naltrexone at Week 8 (n=3,107) | 0.0 (0.0) | 2.9 (11.13)
  Naltrexone at Week 12/ET (n=4,137) | 0.0 (0.0) | 3.0 (12.67)
  6-β-naltrexol at Baseline (n=127,139) | 216.0 (800.32) | 97.5 (300.17)
  6-β-naltrexol at Week 4 (n=3,115) | 0.0 (0.0) | 86.1 (315.42)
  6-β-naltrexol at Week 8 (n=3,107) | 0.0 (0.0) | 48.3 (156.42)
  6-β-naltrexol at Week 12/ET (n=4,137) | 0.0 (0.0) | 55.6 (163.41)

ADVERSE EVENTS:
Time Frame: From the time of informed consent up to and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or 1 participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Open ALO-02 | ALO-02 To Placebo | ALO-02 To ALO-02
Serious Adverse Events (participants affected / at risk) | 3/410 | 2/134 | 5/146
Other Adverse Events (participants affected / at risk) | 186/410 | 26/134 | 41/146
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open ALO-02 (N=410) | ALO-02 To Placebo (N=134) | ALO-02 To ALO-02 (N=146)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Intermittent claudication (Vascular disorders) | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Drug administration error (Injury, poisoning and procedural complications) | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Cholesterosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open ALO-02 (N=410) | ALO-02 To Placebo (N=134) | ALO-02 To ALO-02 (N=146)
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 3
Constipation (Gastrointestinal disorders) | 61 | 3 | 5
Diarrhoea (Gastrointestinal disorders) | 9 | 6 | 8
Nausea (Gastrointestinal disorders) | 84 | 5 | 21
Vomiting (Gastrointestinal disorders) | 37 | 4 | 9
Dizziness (Nervous system disorders) | 24 | 1 | 6
Headache (Nervous system disorders) | 30 | 7 | 2
Somnolence (Nervous system disorders) | 36 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 26 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less